# Johnson & Johnson Vision Care, Inc.

# Clinical Study Protocol

The effects of contact lenses with experimental dye on visual function

Protocol CR-6100

Version: 2.0, Amendment 1.0

Date: 07 June 2018

Investigational Products: senofilcon A with new UV-blocker

Key Words: senofilcon A-based contact lens with new UV-blocker, ACUVUE® OASYS®, senofilcon A, daily disposable, non-dispensing.

### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

#### TABLE OF CONTENTS

| | COL TITLE, NUMBER, VERSION | 6 |
|---|---|---|
| | OR NAME AND ADDRESS | |
| | CAL MONITOR | |
| | ORIZED SIGNATURES | |
| | GE HISTORY | |
| | PSIS | |
| | ONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | |
| 1. IN | TRODUCTION AND BACKGROUND | |
| 1.1. | Name and Descriptions of Investigational Products | |
| 1.2. | Intended Use of Investigational Products | |
| 1.3. | Summary of Findings from Nonclinical Studies | |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | 17 |
| Uti | 1.1. Relevant Literature References and Prior Clinical Data Relevant to ilized Measures: Disability Glare, Discomfort Glare, Photostress Recoveromatic Contrast | ery, and |
| 1.5.<br>Study | | d Clinical |
| _ | 5.1. Relevant Literature References and Prior Clinical Data Relevant oposed Measures: Halos, Starbursts, Two-Point Thresholds | |
| 2. ST | UDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 20 |
| 2.1. | Objectives | 20 |
| 2.2. | Endpoints | 20 |
| 2.3. | Hypotheses | 21 |
| 3. TA | ARGETED STUDY POPULATION | 22 |
| 3.1. | General Characteristics | 22 |
| 3.2. | Inclusion Criteria | 23 |
| 3.3. | Exclusion Criteria. | 23 |
| 3.4. | Enrollment Strategy | 24 |
| 4. ST | UDY DESIGN AND RATIONALE | 24 |
| 4.1. | Description of Study Design | 24 |
| 4.2. | Study Design Rationale | 24 |
| 4.3. | Enrollment Target and Study Duration | 25 |
| 5. TE | ST ARTICLE ALLOCATION AND MASKING | |
| 5 1 | Test Article Allocation | 25 |

| | 5.2. | Masking | 26 |
|---|---|---|---|
| | 5.3. | Procedures for Maintaining and Breaking the Masking | 26 |
| 6. | STU | JDY INTERVENTION | 27 |
| | 6.1. | Identity of Test Articles | 27 |
| | 6.2. | Ancillary Supplies/Products | 27 |
| | 6.3. | Administration of Test Articles | 27 |
| | 6.4. | Packaging and Labeling | 28 |
| | 6.5. | Storage Conditions | 28 |
| | 6.6. | Collection and Storage of Samples | 28 |
| | 6.7. | Accountability of Test Articles | 28 |
| 7. | STU | JDY EVALUATIONS | 29 |
| | 7.1. | Time and Event Schedule | 29 |
| | 7.2. | Detailed Study Procedures | 30 |
| | VIS | IT 1 | 30 |
| | VIS | IT 2 | 47 |
| | FIN | AL EVALUATION | 50 |
| | 7.3. | Unscheduled Visits | 50 |
| | 7.4. | Laboratory Procedures | 51 |
| 8. | SUI | BJECTS COMPLETION/WITHDRAWAL | |
| | 8.1. | Completion Criteria | 52 |
| | 8.2. | Withdrawal/Discontinuation from the Study | 52 |
| 9. | PRI | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 52 |
| 10 | | EVIATIONS FROM THE PROTOCOL | |
| 11 | . S | TUDY TERMINATION | 53 |
| 12 | | ROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | |
| 13 | . A | DVERSE EVENTS | 55 |
| | 13.1. | Definitions and Classifications | |
| | 13.2. | Assessing Adverse Events | 57 |
| | 13.2 | 2.1. Causality Assessment | 57 |
| | 13.2 | | |
| | 13.3. | Documentation and Follow-Up of Adverse Events | |
| | 13.4. | Reporting Adverse Events | |
| | 13.4 | 1.1. Reporting Adverse Events to Sponsor | 59 |
| | 13.4 | 4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorit 60 | ies |

| 13. | .5. | Event of Special Interest | . 60 |
|---|---|---|---|
| 13. | .6. | Reporting of Pregnancy | . 60 |
| 14. | STA | ATISTICAL METHODS | . 61 |
| 14. | .1. | General Considerations | . 61 |
| 14. | .2. | Sample Size Justification. | . 61 |
| 14. | .3. | Analysis Populations | . 61 |
| 14. | .4. | Level of Statistical Significance | . 61 |
| 14. | .5. | Primary Analysis | . 62 |
| 14. | .6. | Secondary Analysis | . 62 |
| 14. | .7. | Other Exploratory Analyses | . 64 |
| 14. | .8. | Interim Analysis | . 64 |
| 14. | .9. | Procedure for Handling Missing Data and Drop-Outs | . 64 |
| 14. | .10. | Procedure for Reporting Deviations from Statistical Plan | . 64 |
| 15. | DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | . 64 |
| 15. | .1. | Electronic Case Report Form/Data Collection | . 64 |
| 15. | .2. | Subject Record | . 65 |
| 16. | DA | TA MANAGEMENT | . 65 |
| 16. | .1. | Access to Source Data/Document | . 65 |
| 16. | .2. | Confidentiality of Information. | . 66 |
| 16. | .3. | Data Quality Assurance | . 66 |
| 17. | MC | NITORING | . 66 |
| 18. | ETI | HICAL AND REGULATORY ASPECTS | . 67 |
| 18. | .1. | Study-Specific Design Considerations | . 67 |
| 18. | .2. | Investigator Responsibility | . 67 |
| 18. | .3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | . 67 |
| 18. | .4. | Informed Consent | . 68 |
| 18. | .5. | Privacy of Personal Data | . 69 |
| 19. | STU | JDY RECORD RETENTION | . 70 |
| 20. | FIN | ANCIAL CONSIDERATIONS | . 70 |
| 21. | PU | BLICATION | . 71 |
| 22. | RE | FERENCES | . 71 |
| APPI | ENDI | X A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | . 73 |
| APPI | ENDI | X B: PATIENT INSTRUCTION GUIDE | . 78 |
| APPI | ENDI | X C: PACKAGE INSERT (APPROVED PRODUCT) | . 79 |

| APPENDIX D: | 82 |
|---|---|
| Lens Fitting Characteristics | |
| SUBJECT REPORTED OCULAR SYMPTOMS/PRO | OBLEMS 90 |
| DETERMINATION OF DISTANCE SPHEROCYLI | |
| BIOMICROSCOPY SCALE | 99 |
| DISTANCE AND NEAR VISUAL ACUITY EVALU | UATION 105 |
| PATIENT REPORTED OUTCOMES | 110 |
| APPENDIX E: DETERMINATION OF EYE DOMINANCY | 112 |
| APPENDIX F: IRIS COLOR | 113 |
| APPENDIX G: SPECTRUM OF THE UV ACTUATOR | 115 |
| APPENDIX H: STARBURST AND HALO IMAGES | 116 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATUR | E PAGE 117 |
| TABLE OF CONTENTS | |
| Figure 1: Study Flowchart | 13 |
| Figure 2: Schematic of the 2-channel Maxwellian optical syst measures. | em used for our dependent |
| Figure 3: Actual Testing System | 37 |
| Figure 4: The xenon (dark line) compared to noon day sun light taken from the NASA solar spectrum measured at the earth's surf | |
| ordinate with respect to the xenon source that will be used in this | |
| Figure 5: Schematic of the dysphotopsia-measuring device | |
| Figure 6: Protototype of testing system for two-point spread func | tions43 |
| Figure 7: Prototype of Testing System for halos and starbursts | |
| TABLE OF CONTENTS | |
| Table 1: Test Articles | 27 |
| Table 2: Ancillary Supplies | |
| Table 3: Time and Events | 29 |

#### PROTOCOL TITLE, NUMBER, VERSION

Title: The effects of contact lenses with new UV-blocker on visual function

Protocol Number: CR-6100

Version: 2.0

Date: 07 June 2018

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR

Name: John R. Buch, O.D., M.S., F.A.A.O. Title: Senior Principal Research Optometrist

Email: jbuch@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, <sup>4</sup> ICH guidelines, <sup>2</sup> ISO 14155, <sup>1</sup> and the Declaration of Helsinki. <sup>3</sup>

| Author/Study | | |
|---|---|---|
| Responsible Clinician | See Electronic Signature Report John R. Buch, O.D., M.S. Sr. Principal Research Optometrist, JJVC | DATE |
| Co-author | | |
| Clinical Operations<br>Manager | | |
| Biostatistician | | |
| Data Management | | |
| Approver | | |
| Reviewer | | |

# **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section | Date |
|---|---|---|---|
| | | Number(s) Affected | |
| 1.0 | John R. Buch | Original Protocol | 28 March 2018 |
| 2.0 | John R. Buch | Update visit windows from 1-14 day to 1-28 | 07 June 2018 |
| | | days | |

# **SYNOPSIS**

| Protocol Title | The effects of contact lenses with experimental dye on visual function |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Development phase 3 |
| Trial Registration | This study will be registered on ClinicalTrials.gov. |
| Test Article(s) | Investigational Products: senofilcon A-based contact lens with new UV blocker. |
| | Control Products: ACUVUE OASYS |
| Wear and Replacement<br>Schedules | Wear Schedule: daily wear Replacement Schedule: daily |
| Objectives | The objective of this study is to objectively measure potential benefits of the new UV blocker. |
| Study Endpoints | Primary endpoint(s): two-point light thresholds, halo and starbursts geometry. Secondary endpoint(s): photostress recovery (PR) time, glare |
| | discomfort threshold (GDc), glare disability threshold (GDs), heterochromatic contrast. |
| | Other observations: on-eye light transmission, ocular physiology, subjective response. |
| Study Design | This is a single-site, two-visit, contralateral, non-dispensing, randomized, controlled and subject-masked study. At Visit 1 subjects will be randomly assigned to wear one of two lens wear sequences (left: Test, right: Control or left: Control, right: Test) and will undergo Psychometric Testing A. |
| | At Visit 2, there are two levels of randomization, first subjects will be assigned randomly to 1 of 2 lens wear sequences (left: Test, right: Control or left: Control, right: Test) and subjects will then be randomized to the order of the Test lens activation (activated/inactivated or inactivated/activated) and will then undergo Psychometric Testing B. |
| | See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1: Study Flowchart). |
| Sample Size | Approximately 66 eligible subjects will be enrolled and randomized into the study. Approximately 60 subjects are targeted to complete the study. Of these, approximately 40 will be in the 18-39 age range, and approximately 20 in the 40-65 age range. |

| Study Duration | There are two study visits that will last approximately 2-3 hours each. At least 24 hours must separate the end of Visit 1 and the beginning of Visit 2. Once enrolled, all subjects are expected to complete both visits within 28 days. The study enrollment period will be approximately 6 weeks. |
|---|---|
| Anticipated Study Population | All subjects will be habitual wearers of spherical soft silicone hydrogel contact lenses that can be fit with the lens powers available for this study. Healthy male and female volunteers of any race and ethnicity will be recruited that are ≥18 and ≤39 years of age (~2/3 of the total sample) and are ≥40 and ≤65 years of age (~1/3 of the total sample). |
| Eligibility Criteria (Inclusion) | <ol> <li>Potential subjects must satisfy all of the following inclusion criteria to be enrolled in the study: <ol> <li>The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.</li> <li>Appear able and willing to adhere to the instructions set forth in this clinical protocol</li> <li>Between 18 and 65 (inclusive) years of age at the time of screening.</li> <li>Be a current spherical soft silicone hydrogel contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week wear time over the last 30 days by self-report.</li> </ol> </li> <li>Inclusion Criteria after Baseline</li> <li>The subject's vertex-corrected spherical equivalent distance refraction must be in the range of -1.00 through -4.50 D in each eye.</li> <li>The subject has a best corrected visual acuity of 20/25 or</li> </ol> |

### Eligibility Criteria Potential subjects who meet any of the following criteria will (Exclusion) be excluded from participating in the study: 1. Currently pregnant or breastfeeding. 2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear. 3. Any autoimmune disease or use of medication, which may interfere with contact lens wear. Habitual medications used by successful soft contact lens wearers are considered acceptable. 4. Entropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or aphakia. 5. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.). 6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear. 7. Multifocal, toric or extended wear contact lens correction. 8. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment. 9. History of binocular vision abnormality or strabismus. 10. Any infectious disease (e.g., hepatitis, tuberculosis) or contagious immunosuppressive diseases (e.g., HIV) by self-report. 11. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician). Exclusion Criteria after Baseline 12. Any ocular infection. 13. Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear. Disallowed Use of any prescription or over-the-counter (OTC) Medications/Interventions medications that may affect contact lens wear from 24 hours prior to receiving the study product through the study period of 2 visits. Habitual medications taken by successful soft contact lens wearers are considered acceptable.

| Measurements and Procedures | The new UV-blocker has the potential to provide visual benefits that go beyond the correction of ametropia. This study will objectively measure these benefits using an optical bench set-up. |
|---|---|
| Microbiology or Other<br>Laboratory Testing | None |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any SAE where relationship to study agent cannot be ruled out, will result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study-<br>Specific Materials | EyeCept preservative-free eyedrops, optical bench set-up. |
| Principal Investigator(s) and Study Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |

Figure 1: Study Flowchart



#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CIE Corneal Infiltrative Event
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

HEV High Energy Visible
IB Investigator's Brochure
ICF Informed Consent Form

ICH International Council on Harmonisation IDE Investigational Device Exemption IEC Independent Ethics Committee IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

MPMVA Maximum Plus to Maximum Visual Acuity

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide
PQC Product Quality Complaint
PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation SKU Stock Keeping Unit

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

UV Ultraviolet VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Photochromic spectacle lenses have been tested for their ability to improve visual functions under intense light conditions.<sup>5</sup> In that study, 75 subjects were tested in a subject-masked cross-over design (a transparent spectacle lens was compared to a partially activated photochromic). Subjects wearing the photochromic lenses (a variety of types were used) showed significant improvements in photostress recovery, glare disability, and glare discomfort. Recently, a similar effect was found for photochromic contact lenses (unpublished) using a contralateral design. Compared to a clear contact in one eye (the OASYS), a photochromic contact demonstrated improved photostress recovery, glare disability and discomfort (and chromatic contrast, an effect not seen as strongly in the parallel photochromic spectacle study). Although compelling as a first study, two major questions remain.

Question 1: Are the deleterious effects of light scatter continuous? Glare disability specifically refers to visual function under intense light circumstances. Light enters the eye, is scattered by the anterior media (or even surface characteristics of the cornea such as excess lacrimal fluid or even contact lenses), and this scatter interferes with visual function (e.g., by veiling an image). Since this scattering, however, is caused by static features of the eye (ranging from the optical quality of a contact lens to in homogeneities within the cornea or lens), it is also present under low light conditions. Stated differently, scattering is no more excessive in intense light, it is just more aversive. Scattering under low-moderate light conditions may not be as bothersome but it is much more pervasive: to wit, it degrades our vision under all lighting conditions.

One very convenient way of measuring the visual effects of low-level light scatter is based on the two-point-light spread technique. Two small points of light are used (simulated sunlight is the best to use for ecological validity). The light can either start as one point (subjects then

determine the minimum distance needed to see two points) or two points (the subjects indicate when only one point is perceived). The intensity of the points can be varied from very high to low. As the point spread function of the eye is increased, the distance between when the points are deemed distinct is also proportionally increased.

Question 2: What aspects of glare are improved by filtering? Glare disability is measured by exposing subjects to a bright source of light and then measuring how this light interferes with some form of visual discrimination (either the glare source can be varied or the intensity of the target). In this scenario, one is simply testing how bright light interferes with some aspect of visual function (such as contrast discrimination). It does not, however, measure how the glare light itself is scattered. For example, light can scatter uniformly causing a homogenous veil (similar to a ganzfeld).<sup>7</sup> It can also spread in what appears like spokes or starbursts (this sometimes referred to as positive dysphotopsia and is caused by high-order aberrations). These appear to be particularly pernicious when individuals have gone through laser correction of myopia and cataract surgery (dysphotopsia is the number one problem following successful cataract surgery, around 51% of patients). They also, however, accompany a plethora of other conditions including dry eye, astigmatism, epiphora, mild-traumatic brain injury, epicanthic eye structure, increased lens density (particularly glycemic), etc. Ritschel et al. (2009) described these autonomous glare phenomenon

"In general the effects of glare can be divided into bloom, a general loss of contrast in the surroundings of the retinal image of the light-source (veil), and flare which comprises the ciliary corona (the sharp needles) and the lenticular halo surrounding the light."

In the previous study, we measured the first aspect of glare (the veil or bloom). In this study, we would like to measure the latter two, the halo and spokes.

#### Practical implications:

Visual disturbance in the form of halos and starbursts is common; when the issues become clinical, they are often referred to as dysphotopsia. Dysphotopsia, for instance, is common in patients who have had LASIK surgery to correct vision. In fact, it has been argued that these complications are why LASIK has dropped by more than 50 percent, from 1.5 million procedures a year in 2007 to 604K in 2015 (e.g., see <a href="lasikcomplications.com">lasikcomplications.com</a>). Dysphotopsia is also common in patients who are progressing from early, pre-cataractous vision toward severe (operable) cataract (about half of the population over 70 years). Dysphotopsia is particularly evident during night time driving and is one of the major reasons why older adult patients stop driving at night. It is also a major reason for displanting IOLs that were implanted to correct cataracts.

It is not simply older patients, however, who have these issues. To demonstrate this (unpublished data), we measured halos and visual starbursts in a sample of young subjects (17-22 years of age). The size of the central halo for these young subjects varied by a factor of six (range = 3-13 cm). Their peripheral spokes varied by nearly a factor of three (6-15). Hence, even in these young healthy and largely homogeneous subjects the range (and aversive ness) was very large. This is why a number of spectacle lenses (even contact lenses, see

http://blog.uniqso.com/contact-lenses-help-reduce-halos-glare/) are specifically marketed for their ability to reduce halos and starbursts.

This study will have one Control lens (ACUVUE OASYS), and one Test lens (Investigational). However, the one Test lens will be evaluated under two separate lighting conditions making three study articles altogether.

#### 1.1. Name and Descriptions of Investigational Products

This study will evaluate the Test lens vs. the Control lens. The Test lens is senofilcon A with a new UV blocker, while the Control lens is senofilcon A without the new UV blocker (i.e., ACUVUE OASYS). Further details about the test articles are found in Section 6 of this protocol.

#### 1.2. Intended Use of Investigational Products

The intended use of the investigative product in this study is for correcting myopia and for the attenuation of bright lights. The study articles will be worn contralaterally in a daily wear, daily disposable modality for approximately 2 hours on both days of the study. The study articles will not be dispensed.

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding the senofilcon A-based contact lens with new UV blocker, refer to the latest version of the Investigator's Brochure

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

In addition to the correction of their myopia, subjects are likely to experience a reduction of bright lights.

For the most comprehensive risk and benefit information regarding the senofilcon A-based contact lens with new UV blocker, refer to the latest version of the Investigator's Brochure.

# 1.4.1. Relevant Literature References and Prior Clinical Data Relevant to Previous Utilized Measures: Disability Glare, Discomfort Glare, Photostress Recovery, and Chromatic Contrast

- Colombo, L., Melardi, E., Ferri, P., Montesano, G., Attaalla, S. S., Patelli, F., ... & Rossetti, L. (2017). Visual function improvement using photocromic and selective blue-violet light filtering spectacle lenses in patients affected by retinal diseases. BMC ophthalmology, 17(1), 149.
- Huang, W. J., Yang, Y., & Luo, M. R. (2017). Discomfort glare caused by white LEDs having different spectral power distributions. Lighting Research & Technology, 1477153517704996.
- Lee, H. S., Kim, J. Y., Subramaniyam, M., Park, S., & Min, S. N. (2017). Evaluation of quantitative glare technique based on the analysis of bio-signals. Ergonomics, 60(10), 1376-1383.

- Longley, C., & Whitaker, D. (2016). Google Glass Glare: disability glare produced by a head-mounted visual display. Ophthalmic and physiological optics, 36(2), 167-173.
- Mahjoob, M., Heydarian, S., & Koochi, S. (2016). Effect of yellow filter on visual acuity and contrast sensitivity under glare condition among different age groups. International ophthalmology, 36(4), 509-514.
- Mehri, A., Farhang Dehghan, S., Hajizadeh, R., Zakerian, S. A., Mohammadi, H., & Abbasi, M. (2017). Survey of discomfort glare from the headlamps of cars widely used in Iran. Traffic injury prevention, (just-accepted).
- Pierson, C., Bodart, M., Cauwerts, C., & Wienold, J. (2017). Discomfort glare from daylighting: study of factors influencing discomfort glare perception and validation of a universal discomfort glare index. In VELUX Daylight Symposium.
- Pierson, C., Wienold, J., & Bodart, M. (2017). Discomfort glare from daylighting: influence of culture on discomfort glare perception. In CIE 2017 Midtern Meeting.
- Ritschel, T., Ihrke, M., Frisvad, J. R., Coppens, J., Myszkowski, K., & Seidel, H. P. (2009). Temporal Glare: Real-Time Dynamic Simulation of the Scattering in the Human Eye. In Computer Graphics Forum 28, 2, 183-192.
- Rodriguez, R. G., Yamín Garretón, J. A., & Pattini, A. E. (2016). Glare and cognitive performance in screen work in the presence of sunlight. Lighting Research & Technology, 48(2), 221-238.
- Rosli, S. A., Aladin, A. Z., Muhamad, N., & Chen, A. H. (2016). Comparison of visibility threshold on different chromatic contrast objects. Social and Management Research Journal, 13(1), 106-115.
- Sewall, A. A. S., Borzendowski, S. A. W., Tyrrell, R. A., Stephens, B. R., & Rosopa, P. J. (2016). Observers' Judgments of the Effects of Glare on Their Visual Acuity for High and Low Contrast Stimuli. Perception, 45(7), 755-767.
- Siah, W. F., O'Brien, C., & Loughman, J. J. (2017). Macular pigment is associated with glare-affected visual function and central visual field loss in glaucoma. British Journal of Ophthalmology, bjophthalmol-2017.
- Stringham, J. M., O'Brien, K. J., & Stringham, N. T. (2016). Macular carotenoid supplementation improves disability glare performance and dynamics of photostress recovery. Eye and Vision, 3(1), 30.
- Wahl, S., Fornoff, L., Ochakovski, G. A., & Ohlendorf, A. (2017). Disability glare in soft multifocal contact lenses. Contact Lens and Anterior Eye.

See also the Investigator's Brochure.<sup>9</sup>

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

evaluated the same study lenses as the current study on a similar optical bench set up. In that study, the Test and Control lenses were subjected to a 395 nm light source that would normally be present in the outdoor environment on a sunny day. The Test lens performed better than the Control lens in this simulated environment. However, previous studies have shown an indoor benefit of the Test lens over the Control lens and this remains unexplained - particularly since indoor light is typically absent of any significant 395 nm light. It is important to understand whether the same optical bench metrics

(photostress recovery, discomfort glare, disability glare, and heterochromatic contrast) can help explain the indoor benefit.

The same previous studies that have shown an indoor benefit with the Test lens have shown a benefit with daytime and nighttime driving. Subjects typically report that their vision is better and they have less issues with bright lights. The mechanism behind this remains unexplained. The current study will investigate this area by evaluating the magnitude of dysphotopsia with the Test and Control lens under simulated daytime and nighttime wavelengths.

# 1.5.1. Relevant Literature References and Prior Clinical Data Relevant to New Proposed Measures: Halos, Starbursts, Two-Point Thresholds

- Artal, Pablo, and Rafael Navarro (1992). Simultaneous measurement of two-point-spread functions at different locations across the human fovea. Applied optics 31.19: 3646-3656.
- Aujla, M., Wolffsohn, J. S., & Sheppard, A. L. (2015). Halo size and subjective complaints of dysphotopsia in a normal population. Investigative Ophthalmology & Visual Science, 56(7), 4314-4314.
- Babizhayev, M. A., Minasyan, H., & Richer, S. P. (2009). Cataract halos: a driving hazard in aging populations. Implication of the Halometer DG test for assessment of intraocular light scatter. Applied ergonomics, 40(3), 545-553.
- Brown, S. M. (2004). Measuring starbursts. Journal of Cataract & Refractive Surgery, 30(12), 2646-2647.
- Davison, J. A. (2000). Positive and negative dysphotopsia in patients with acrylic intraocular lenses. Journal of Cataract & Refractive Surgery, 26(9), 1346-1355.
- De Boer, J. B. (1967). Visual perception in road traffic and the field of vision of the motorist. In Public Lighting (pp. 11-96).
- Finney, D. J. (1971). Probit analysis (3rd ed.). Cambridge: University Press.
- Gowrisankaran, S., Sheedy, J. E., & Hayes, J. R. (2007). Eyelid squint response to asthenopia-inducing conditions. Optometry and Vision Science, 84, 611-19.
- Hammond, B. R. (2012). The visual effects of intraocular filters. Scientifica, 2012. doi:10.6064/2012/424965
- Hammond, B. R., Bernstein, B., & Dong, J. (2009). The effect of the AcrySof Natural lens on glare disability and photostress. American Journal of Ophthalmology, 148(2), pp. 272-276.
- Hammond, B. R., Renzi, L. M., Sachak, S., & Brint, S. F. (2010). Contralateral comparison of blue-filtering and non-blue-filtering intraocular lenses: glare disability, heterochromatic contrast, and photostress recovery. Clinical Ophthalmology, 4, pp. 1465-1473.
- Kenward, M. G., & Roger, J. H. (1997). Small sample inference for fixed effects from restricted maximum likelihood. Biometrics, 53(3), pp. 983-997.
- Mecherikunnel, A. T., & Richmond, J. C. (1980). Spectral distribution of solar radiation.
   Technical Memorandum 82021, NASA, Goddard Space Flight Center, Greenbelt, Maryland.
- Nahar, N. K., Sheedy, J. E., Hayes, J., & Tai, Y. C. (2007). Objective measurements of lower-level visual stress. *Optometry and Vision Science*, 84(7), 620-629.
- Renzi, L. and Hammond, B.R. (2016). The effects of photochromic lenses on visual performance. Clinical and Experimental Optometry, 1-7.

- Ritschel, T., Ihrke, M., Frisvad, J. R., Coppens, J., Myszkowski, K., & Seidel, H. P. (2009, April). Temporal Glare: Real-Time Dynamic Simulation of the Scattering in the Human Eye. In Computer Graphics Forum (Vol. 28, No. 2, pp. 183-192). Blackwell Publishing Ltd.
- Sayre, R. M., Cole, C., Billhimer, W., Stanfield, J., & Ley, R. D. (1990). Spectral comparison of solar simulators and sunlight. Photodermatol Photoimmunol Photomed, 7, pp. 159-165.
- Sheedy, J. E., Truong, S. D., & Hayes, J. R. (2003). What are the visual benefits of eyelid squinting?. *Optometry and vision science*, 80(11), 740-744.
- Stringham, J. M., Fuld, K., & Wenzel, A. J. (2003). Action spectrum for photophobia. *JOSA A*, 20(10), 1852-1858.
- Valverde, J. A., & Gonza, R. (2003). Simple device for quantifying the influence of halos after lasik surgery. Journal of biomedical optics, 8(4), 663-667.
- Westheimer, G. (1975). Visual acuity and hyperacuity. Investigative Ophthalmology, 14(8), pp. 570-572.

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

#### Primary Objective(s)

The primary objective of this study is to investigate the daytime and nighttime driving benefit seen with previous studies. It will determine whether the Test lens can demonstrate an objective benefit in the absence and presence of a UV/HEV light source over the Control lens. The size of dysphotopsia (halos, starburst, scattering) will be measured.

#### Secondary Objective(s)

The secondary objective of this study is to investigate the indoor benefit seen with previous studies. It will determine whether the investigational lens can demonstrate an objective benefit in the absence of a UV/HEV light source over the Control lens. Psychophysical measures such a photostress recovery, disability glare, discomfort glare, and chromatic contrast will be used.

#### Exploratory Objective(s)

The on-eye light transmission will be measured on a sampling of subjects by measuring absolute sensitivity to test lights with activated and inactivated lenses. Slit lamp findings and subjective ratings will be monitored.

#### 2.2. Endpoints

There is one Control lens and one Test lens in this study. However, the Test lens is evaluated with and without an added UV/HEV light source. The testing conditions and endpoints are summarized here with detail provided.

| Visits | Compare | | Endpoints | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Lens | Photo | Disabil | Discom | CC | Halo | Starb | Scatt |
| 1 | A/B | ✓ | ✓ | ✓ | ✓ | - | - | - |
| 2 | A/B<br>A/C | - | - | - | 1 | <b>√</b> | ✓ | <b>√</b> |

- A: Control lens, B: investigational lens without added UV/HEV light, C: investigational lens with added UV/HEV light
- Photo: photostress recovery, Disabil: disability glare, Discom: discomfort glare, CC: chromatic contrast,
   Halo: haloes, Starb: starbursts, Scatt: scattering

#### Primary Endpoint(s)

Positive dysphotopsia can take many forms and can manifest itself as scintillating vision (scattering), seeing arcs, flare, flashes, starbursts and haloes. The investigational lens has the potential to decrease these symptoms, particularly in the presence of an added UV/HEV light source. In this study, the investigators will evaluate the degree of light scattering, haloes, and starbursts using a two-point light threshold test and a newly-designed halometer. Light scattering, halos, and starbursts are more obvious at night prompting testing to occur with an inactivated lens. However, they are also present during the day prompting testing to also occur with an activated lens.

#### Secondary Endpoint(s)

The psychophysical metrics of photostress recovery, disability glare, discomfort glare, and chromatic contrast will be recorded in the absence of an added UV/HEV light source. An optical bench set up will be used. This will relate to indoor vision when the lenses are less likely to be activated.

#### Other Exploratory Endpoint(s)

Knowing the light transmission through the contact lenses is of particular interest to the development team. A sampling of subjects will undergo additional absolute sensitivity testing to estimate the in vivo light transmission. Slit lamp findings and subjective ratings will be monitored.

#### 2.3. Hypotheses

Primary Hypotheses (each is considered independent)

- 1. Light Scattering
  - a. The Test lens (in the <u>absence</u> of an additional UV/HEV light source) will be statistically lower than the Control lens with respect to light scattering as measured using the two-point light threshold instrument.
  - b. The Test lens (in the <u>presence</u> of an additional UV/HEV light source) will be statistically lower than the Control lens with respect to light scattering as measured using the two-point light threshold instrument.

#### 2. Haloes

- a. The Test lens (in the <u>absence</u> of an additional UV/HEV light source) will be statistically lower than the Control lens with respect to halos. This is measured using the halometer instrument.
- b. The Test lens (in the <u>presence</u> of an additional UV/HEV light source) will be statistically lower than the Control lens with respect to halos. This is measured using the halometer instrument.

#### 3. Starbursts

- a. The Test lens (in the <u>absence</u> of an additional UV/HEV light source) will be statistically lower than the Control lens with respect starbursts as measured using the halometer instrument.
- b. The Test lens (in the <u>presence</u> of an additional UV/HEV light source) will be statistically lower than the Control lens with respect starbursts as measured using the halometer instrument.

#### Secondary Hypotheses (each is considered independent)

- 1. The Test lens (in the absence of an additional UV/HEV light source) will be statistically lower than the Control lens with respect to photostress recovery time (seconds) as measured using the optical bench instrument.
- 2. The Test lens (in the absence of an additional UV/HEV light source) will be statistically higher than the Control lens with respect to disability glare threshold as measured using the optical bench instrument.
- 3. The Test lens (in the absence of an additional UV/HEV light source) will be statistically lower than the Control lens with respect to discomfort glare (eyelid squinting) as measured using the optical bench instrument.
- 4. The Test lens (in the absence of an additional UV/HEV light source) will be statistically higher than the Control lens with respect to chromatic contrast threshold than as measured using the optical bench instrument.

#### Other Hypotheses

1. In vivo light transmission will be collected on a sampling of subjects for informational purposes only. Slit lamp findings and subjective ratings will be described describely.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Male and female volunteers of any nationality that satisfy the inclusion and exclusion criteria.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

#### Inclusion Criteria after Screening

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol
- 3. Between 18 and 65 (inclusive) years of age at the time of screening.
- 4. Be a current spherical soft silicone hydrogel contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week wear time over the last 30 days by self-report.

#### Inclusion Criteria after Baseline

- 5. The subject's vertex-corrected spherical equivalent distance refraction must be in the range of -1.00 through -4.50 D in each eye.
- 6. The subject has a best corrected visual acuity of 20/25 or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

#### Exclusion Criteria after Screening:

- 1. Currently pregnant or breastfeeding.
- 2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
- 3. Any autoimmune disease or use of medication, which may interfere with contact lens wear. Habitual medications used by successful soft contact lens wearers are considered acceptable.
- 4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or aphakia.
- 5. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
- 6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
- 7. Multifocal, toric or extended wear contact lens correction.
- 8. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
- 9. History of binocular vision abnormality or strabismus.
- 10. Any infectious disease (e.g., hepatitis, tuberculosis) or contagious immunosuppressive diseases (e.g., HIV) by self-report.
- 11. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).

#### Exclusion Criteria after Baseline

- 12. Any ocular infection.
- 13. Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

The study is a single-site, controlled, randomized, subject-masked, non-dispensing, contralateral design. The study begins with an initial visit (Visit 1 - Day 0), if a subject is found to meet all eligibility criteria, then they will be randomized to one of two lens wear sequences (Left: Test, Right: Control or Left: Control, Right: Test); otherwise a subject will be deemed ineligible for this study.

If a subject is found eligible and was 'dispensed' study lenses at the initial visit, then one additional visit will occur. Visit 2 will occur no sooner than 24 hours after Visit 1 and no later than 28 days after visit 1. Each visit will last approximately 2-3 hours each. Unscheduled visits may occur during the course of the study.

#### 4.2. Study Design Rationale

This study will be executed using a contralateral design. There are several benefits to this choice of design. First, we intend to relate performance with the investigational lens in its activated and inactivated states to baseline light sensitivity. A contralateral design will allow us to compare performance with both activation states within the same individual, ostensibly with the same baseline light sensitivity. Second, other subject factors that can influence visual performance, such as iris color and absorption of test lights via macular pigment, are better controlled using this design. Third, in psychophysical testing, which is the gold standard for many of the visual functions being tested, participants make judgments about some event threshold, such as when an image disappears or how large or bothersome or intense a visual event appears. Participants may have different criteria for threshold events that are internally consistent within subjects but can vary between subjects. A contralateral design allows the investigational lens to be compared within subjects, with consistent criteria for threshold events. Given the fact that sufficient time will be taken between measures, in some cases 24 hours or more, carryover effects are unlikely.

#### 4.3. Enrollment Target and Study Duration

Approximately 66 subjects will be enrolled to complete approximately 60 at a single site. The point of study enrollment is the execution and completion of the signed Informed Consent document. Subjects will be stratified into one of two age groups using a 2:1 allocation ratio:

- 40 subjects ±3 in age group 18-39
- 20 subjects ±3 in age group 40-65

There are two study visits that will last approximately 2-3 hours each. At least 24 hours must separate the end of Visit 1 and the beginning of Visit 2. Once enrolled, all subjects are expected to complete both visits within 28 days. The study enrollment period will be approximately 6 weeks.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

Use of the test articles will be randomized using a randomization scheme supplied by the study biostatistician.

This is a single-site, two-visit, contralateral, subject-masked, non-dispensing and randomized study. The study lenses will be worn in a contralateral and random fashion. At visit 1, a block size of (2) sequences will be used to randomly assign subjects to one of two lens wear sequences (Left: Test, Right: Control or Left: Control, Right: Test).

At visit 2, there are two levels of randomization, a block size of (2) sequences will be used to randomly assign subjects to one of two lens wear sequences (Left: Test, Right: Control or Left: Control, Right: Test). Once subjects are randomized to a lens wear sequence, subjects will then be randomized to the order of Test lens activation (activated/inactivated or inactivated/activated).

The random scheme for each visit will be generated by site using the PROC PLAN procedure from SAS Software Version 9.4 or higher (SAS Institute, Cary, NC).

The study site must follow the randomization scheme provided and complete enrollment according to the randomization list and not pre-select or assign subjects. The randomized assignment of subjects will be performed at the first visit prior to the first fitting. The following must have occurred prior to randomization:

- Informed consent has been obtained
- Subject meets all the inclusion / exclusion criteria
- Subject history and baseline information has been collected

#### 5.2. Masking

This is a subject-masked study. Masking will be used to reduce potential bias. Subjects will be unaware of the identity of the investigational product. Investigators and clinical site personnel involved in the data collection will not be masked as to the identity of the investigational product. Although the subjects will not be aware of which study lens is going on which eye, the dynamic nature of the test lens during the assessments may give the identity.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued will be replaced.

#### 5.3. Procedures for Maintaining and Breaking the Masking

The identity of the study lenses will be masked to the subjects by over labeling the blister pack of the study lens. The label will contain the study number, lot number, sphere power, expiration date and the randomization codes S and N.

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

**Table 1: Test Articles** 

| | Test | Control |
|---|---|---|
| Name | ECL100 | ACUVUE OASYS |
| Manufacturer | JJV | JJV |
| Lens Material | senofilcon A | senofilcon A |
| Nominal Base Curve @ 22 °C | 8.4 | 8.4 |
| Nominal Diameter @ 22 °C | 14.0 | 14.0 |
| Nominal Distance Powers (D) | -1.00 through -4.50 | -1.00 through -4.50 |
| Water Content (Optional) | 38 | 38 |
| Center Thickness (Optional) | 0.085 | 0.070 |
| Oxygen Permeability (Dk) | 103 | 103 |
| Wear Schedule in Current Study | Daily | Daily |
| Replacement Frequency | Daily | Daily |
| Packaging Form (vial, blister, etc.) | Blister | Blister |
| Other distinguishing items (e.g., dye, packaging solution, optical design, etc.) | New UV/HEV<br>blocker | NA |

Approximately 25 lenses per stock keeping unit (SKU) will be provided based on 66 subjects, 2-periods, contralateral, non-dispensing design, US population normalized for peak SKUs and a safety factor of 50%.

#### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

**Table 2: Ancillary Supplies** 

| | Solution |
|---------------------------|-------------------------|
| Solution Name/Description | EyeCept Rewetting Drops |
| Manufacturer | Optics Laboratories |
| Preservative | NA |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

#### 6.4. Packaging and Labeling

The test articles will be packaged in blisters as the primary packaging. The test article will be over-labeled to mask the subject to the identity of the lens. The test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:



### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions and stored out of direct sunlight or other source of UV/HEV radiation.

#### 6.6. Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused

#### 3. The number and reason for unplanned replacements

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles, and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

Site Instructions for Test Article Receipt and Test Article Accountability for additional information.

#### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1 | Visit 2 |
|---|---|---|
| | Screening, Baseline 1, | Baseline 2, |
| | Psychometric Testing A | Psychometric Testing B |
| Time Point | Day 1 | 1-28 Days after Visit 1 |
| Estimated Visit Duration | 2.5 hours | 2.5 hours |
| Statement of Informed Consent | X | |
| Demographics | X | |
| Medical History/Concomitant | x | x |
| Medications | X | A |
| Habitual Contact Lens Information | X | |
| Inclusion/Exclusion Criteria | X | |
| Baseline Questionnaires | X | |
| Entrance Visual Acuity | X | X |
| Subjective Sphero-Cylindrical | | |
| Refraction | X | |
| Slit Lamp Biomicroscopy | X | X |
| Lens Selection | X | X |
| Lens Insertion & Settling | X | X |
| Visual Acuity and Over Refraction | X | X |
| Lens Power Modification (if | x | x |
| applicable) | A | A |
| Subject Reported Ocular Symptoms | X | X |
| Lens Fit Assessment | X | X |
| Snellen Distance Visual Acuity | X | X |
| Study Assessments (dysphotopsia and/or psychophysical testing) | X | х |

| Visit Information | Visit 1 | Visit 2 |
|---|---|---|
| | Screening, Baseline 1, | Baseline 2, |
| | Psychometric Testing A | Psychometric Testing B |
| Time Point | Day 1 | 1-28 Days after Visit 1 |
| Estimated Visit Duration | 2.5 hours | 2.5 hours |
| Post-assessment Questionnaire | X | X |
| Study Completion | | X |

# 7.2. Detailed Study Procedures

VISIT 1

Subjects must enter Visit 1 wearing their own contact lenses.

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign<br>the Statement of Informed Consent before<br>being enrolled into the study. The Principal<br>Investigator or his/her designee conducting<br>the informed consent discussion must also<br>sign the consent form. |
| | | Note: The subject must be provided a signed copy of this document. |
| 1.2 | Demographics | Record the subject's year of birth, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. |
| 1.5 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after screening, proceed to Final Evaluation and |
| | | complete Subject Disposition. Refraction and<br>Biomicroscopy forms are not required. |

| | Visit 1: Baseline | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.6 | Baseline<br>Questionnaire | In order to determine how light sensitive participants in the study are at baseline, participants will be administered several questions from various validated instruments that measure self-reported light sensitivity. | |
| 1.7 | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual contact lens correction in place. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |
| 1.8 | Remove Habitual<br>Lens | If applicable, the subject's habitual contact lenses will be removed and stored in their own lens case. If they forgot to bring their lens case, one will be provided to them. | |
| 1.9 | Subjective Sphero-<br>cylindrical<br>Refraction | Perform subjective best sphere refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use a balancing technique (e.g., the duochrome test for binocular balancing, or the binocular blur balancing test, etc.,) and record the best corrected distance visual acuity (OD, OS, and OU) to the nearest letter. | |
| 1.10 | Eye Dominancy | The investigator will determine eye dominancy of the subject by first using the +1.00 blur test. If this fails to determine dominancy, then the sighting test will be used. See Appendix E. | Appendix<br>E |
| 1.11 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If any of these slit lamp findings are grade 3 or higher, the subject may not continue at this time, but may return up to one additional time to determine eligibility. If discontinued a final examination must be completed. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. | |

| Visit 1: Baseline | | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.12 | Iris Color | The investigator will record the subject's iris color based on the scale provided (Appendix F). | Appendix F |
| 1.13 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after two baseline attempts at Visit 1, proceed to Final Evaluation and complete all forms. | |
| 1.14 | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on the refraction. Record the test condition. | |
| 1.15 | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Replace damaged lenses if applicable. | |
| 1.16 | Lens Settling 1 | Allow the study lenses to settle for a minimum of 5 minutes. | |
| 1.17 | Subjective Best<br>Sphere Over<br>Refraction | Perform subjective best sphere refraction over the study lenses (adopt the maximum plus to maximum visual acuity (MPMVA) approach. | |
| 1.18 | Lens Power<br>Modification (if<br>applicable) | Adjust the lens power if the subject's best sphere over-refraction is not plano. For any power modification, repeat steps (1.15-1.17). One power modification is allowed. | |
| 1.19 | Lens Settling 2 | Please wait a total of 10 minutes from final lens insertion to continue. | |
| 1.20 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.21 | Visual Acuity | Record the best corrected Snellen <u>distance</u> visual acuity to the nearest letter (OD and OS). Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 1.22 | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: • limbal exposure at primary gaze or with extreme eye movement |
| | | <ul> <li>edge lift</li> <li>excessive movement in primary and up gaze</li> <li>insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up</li> <li>Note: if lens fit is unacceptable subject will be discontinued from the study.</li> </ul> |
| 1.23 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Visual acuity is 20/30 or better OD and OS 2. The lens fit is acceptable OD and OS 3. Investigator approval. If the Investigator does not approve the wearing of the study lenses for the psychophysical testing, then the study is terminated for that subject. |
| 1.24 | Lenses Worn in<br>Clinic | The lenses will be released for approximately two hours. 1. The subjects must wear both study lenses the entire time. 2. The lenses will be worn as daily wear only. 3. Rewetting drops are permitted if needed. |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| | | Note: In the event a lens is lost or damaged, it will be replaced immediately. Note: A clinic-only-wear Patient Instruction Guide will be provided. |
| 1.25 | Psychophysical<br>Testing Sequence | At Visit 1, all subjects will proceed to Psychophysical Testing A: This includes photostress recovery, discomfort glare, disability glare, and heterochromatic contrast in the absence of an activating light source. Following the psychometric testing by the co-investigator, the subject will return to the principal investigator to complete the study visit as described in steps 1.26-1.28. |
| 1.26 | Lens Removal | The worn study lenses will be removed and discarded. |
| 1.27 | Exit Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. Ocular adverse events shall be those that grade 3 or 4 on the FDA scale. The study monitored must be notified immediately. The AE will be followed to resolution at which time the subject will be terminated from the study. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 1.28 | Exit VA | Record subjects' distance Snellen visual acuity, OD, OS, and OU to the nearest letter with their habitual correction in place (spectacles or contact lenses). Schedule Visit 2 at least 24 hours and no more than 28 days from now. |

#### Psychophysical Testing A: Photostress / Glare / Chromatic Contrast

#### **Apparatus**

Four efficacy parameters will be measured (heterochromatic contrast threshold (HCT), photostress recovery [PR] time, glare disability [GDs], and glare discomfort [GDc]). All tests will utilize the same apparatus, modified for each parameter. The apparatus used to measure HCT, GDs, GDc, and PR is a two-channel Maxwellian view system and is shown in Figure 2 and Figure 3.

The glare source (annulus/disk) and the visual target will be produced by a 1000 Watt xenon arc point source lamp, with a modified housing that allows dual-channel exit (Newport Optics; Irvine, CA). Alignment of the subject's eye with the optical system will be maintained with a forehead rest and a dental impression bite bar that will be custom-fit for each subject. An auxiliary optical channel with a high-resolution camera and monitor will be used to monitor the pupil during testing to ensure proper fixation and sustained alignment, and will be used to measure GDc. The same apparatus, with small variations, will be used to test HCT, GDs, and PR.

All photometric calibrations will be performed using a PR-650 SpectraScan Colorimeter (Photo Research, Inc., Chatsworth, CA). Wedge and neutral density radiometric calibrations will be performed by using a Graseby Optronics United Detection Technology (UDT) instrument (Orlando, FL). The same UDT instrument will be used before every experimental session to ensure that the total light output of the optical system remains constant and consistent throughout the study. The PR-650 can make measurements down to about 380 nm. An additional radiometer (General Tools and Instruments; New York, NY) will be used to measure output farther down into the UV portion of the spectrum.

#### **Investigational contact lenses**

The Investigational lenses will be tested without an additional UV/HEV light source.

#### The test target

The visual target will be the same in all the visual function tests (HCT, GDc, GDs, PR).

#### The background

The background channel will be manipulated to produce either an annulus (for GDs) or a three-degree background field (for GDc and PR). For the HCT test, the same three-degree background will be filtered through a 460 nm interference filter (half-power bandwidth = 8 nm; Edmund Optics; Barrington, NJ) in order to produce a monochromatic field. Xenon was selected as the light source because it has the characteristic broad band emission spectrum (as assessed by the SpectraScan colorimeter) with a CIE chromaticity of u' = 0.25, v' = 0.53. Xenon is widely regarded as a good match for sunlight. For example, in a study of 26 solar simulators, <sup>12</sup> the authors noted that xenon-arc light sources match the most accurately. The xenon spectrum that will be produced by this system is shown in Figure 4 as compared to mid-day sunlight.






Figure 4: The xenon (dark line) compared to noon day sun light (red line). The line in red is taken from the NASA solar spectrum measured at the earth's surface <sup>13</sup> and adjusted along the ordinate with respect to the xenon source that will be used in this study.

| Psychophysical Testing A: Photostress / Glare / Chromatic Contrast | | |
|---|---|---|
| Т | The psychophysical tests described in Steps 1-4 below may occur in any order. No additional UV/HEV activation light source will be used. | |
| Step | Procedure | Details |
| 1 | Glare Disability<br>(GDs) | The target stimulus will be presented for 2 seconds on and 1 second off to reduce the chances that subjects will habituate to the stimulus. A second channel will provide an annulus with an approximately 11-degree inner diameter and 12-degree outer diameter, as shown below. |
| | | Before each trial, the annulus will be set at a level well below that which would cause the target stimulus to be veiled. The experimenter will then adjust, via the neutral-density wedge, the intensity of the annulus until the target stimulus is no longer visible. Participants will indicate that the target has been veiled by pressing a buzzer. |
| | | The experimenter increases the intensity of light scattering within the subjects' test eyes until they cannot effectively see. Unlike the photostress bleach which is set and standard, the intensity is varied in this test, and hence, so is the aversiveness of the dependent variable. This measurement has been conducted successfully, repeatedly, in the past <sup>14</sup> |
| 2 | Heterochromatic<br>Contrast<br>Threshold<br>(HCT) | Chromatic contrast will be measured as thresholds to a variable wavelength central target presented on a short-wave (460 nm) sky-light background. This aspect of the testing is mostly exploratory to see how the contacts influence chromatic contrast. The relation to filtering is very strong as long as there is differential filtering between the target and the background. Light Incident I |

## Psychophysical Testing A: Photostress / Glare / Chromatic Contrast Photostress To measure PR time, participants are exposed to the same target 3 Recovery (PR) used in each of the other visual function tests. participant is comfortably viewing the target, the experimenter will cover the target with a bright, bleaching light. Exposure to the light will cause participants to momentarily lose sight of the target, which will be covered by an afterimage. As the afterimage fades, participants will gradually be able to re-gain sight of the target. PR time will be recorded as the time it takes following exposure to the bleaching light to regain sight of the target. 0 4 Glare Glare discomfort (GDc) will be quantified using the squint Discomfort response and a questionnaire. The discomfort that accompanies (GDc) exposure to light in excess of an individual's adaptive state is accompanied by contraction of the extraocular muscles (squint). The squint response has been shown to be a valid objective indicator of glare discomfort. 15-17 procedure was described bv Gowrisankaran. 18 Degree of squint is calculated as the ratio of the height of the palpebral fissure under normal lighting conditions compared to maximal squint produced during the photostress exposure. A high-resolution camera (AmScope MU300 digital camera; Irvine, CA) will be used and calibrated against a spatial standard before the start of each day of testing. The resultant videos will be analyzed as still frames using AmScope measurement software (Irvine, CA). To determine subjective ratings of GDc, subjects will be asked to rate the degree of discomfort of the photostressor using a single-item questionnaire OD and OS: How bothersome was the glare that you just experienced? Subjects will have the following response options: Extremely bothersome, Very bothersome, Somewhat bothersome, A little bothersome, Not at all

bothersome.

### Psychometric Testing B: Dysphotopsia Evaluation

## **Apparatus**

Three efficacy parameters will be measured (two-point light spread functions, halos, starbursts) for three lens conditions (OASYS, investigational lens without additional UV/HEV light source, investigational lens with additional UV/HEV light source). All tests will utilize the same apparatus, modified for each parameter.

The general optical apparatus is shown in Figure 6 and Figure 7.

The light source will be produced by a 250 Watt xenon arc point source lamp. Alignment of the subject's eye with the optical system will be maintained with a forehead and chin rest assembly. All photometric calibrations will be performed using an ILT 950 (Peabody, MA). and a Graseby Optronics United Detection Technology (UDT) instrument (Orlando, FL). The same UDT instrument will be used before every experimental session to ensure that the total light output of the optical system remains constant and consistent throughout the study. The PR-650 can make measurements down to about 380 nm. An additional radiometer (General Tools and Instruments; New York, NY) will be used to measure output farther down into the UV portion of the spectrum.

## Investigational contact lenses

The investigational lenses will be tested with an additional UV/HEV light source as one of the test conditions. "Activation" will be achieved using an ultraviolet activator consisting of LEDs waveband 365-400 nm that combines with the primary optical path of the system, after the final lens of the optical system (see Figure 7). The spectral output of the ultraviolet LEDs is given in Appendix G. The ultra-violet LEDs will be used, at a low constant rate, while the visual measures (halos, etc.) are being collected. The overall energy at the plane of the eye is  $64~\mu \text{w/cm2}$  (measured using the ILT 950, the graph in Appendix G is the light source at the energy we plan to use during the measurement). As a comparison, the UV activator emits 0.07 mw/cm2 whereas mid-day sunlight measured 11 mw/cm2 using the same instrument (1:00 PM, partially cloudy day, September 18, 2017, Athens, GA using a UVA light meter: General UV254SD).







## Psychometric Testing B: Dysphotopsia Evaluation

The psychophysical tests described in Steps 1-3 below may occur in any order. All three tests will performed twice: once with an UV/HEV activating light source and once with no activating light source. The order of light source testing will be randomized.

| | activating light source. The order of light source testing will be randomized. | |
|---|---|---|
| Step | Procedure | Details |
| 1 | Two-point Light<br>Spread Function | These thresholds are defined as the minimum distance that two points of light are completely distinct. An ascending and a descending method of limits will be used. This measurement takes about 10-15 minutes. Record values OD and OS, in mm (2 decimal places). |
| 2 | Starburst | This is defined as the diameter of the light's lateral spread. Subjects will have the nature of starbursts explained using visual aids prior to the experiment. The investigator will adjust a calibrated custom-made micrometer (two sides with reverse threading) to spread two posts out from a central mid-point. Those posts will be used to define the outer boundaries of the starburst image. Ascending and descending methods of limits would be used based on subject feedback. This measurement takes about 10-15 Calipers are adjusted until the inner edges are just touching the edges of the starburst pattern. minutes. Record values OD and OS, in mm (2 decimal places). Subjects will respond to a single-item post-starburst questionnaire OD and OS: |
| | | How severe / intense was the starburst that you experienced? Subjects will have the following response options: Severe, moderate, mild, not at all. |

# Psychometric Testing B: Dysphotopsia Evaluation

The psychophysical tests described in Steps 1-3 below may occur in any order. All three tests will performed twice: once with an UV/HEV activating light source and once with no activating light source. The order of light source testing will be randomized.

| | 2 2 | The order of light source testing will be randomized. |
|---|---|---|
| Step | Procedure | Details |
| 3 | Halos | Subjects will have the nature of halos explained using visual aids prior to the experiment. The halo measurement will utilize the same light source as the starburst and two-point measures to produce the halo. The same calibrated micrometer from the starburst test will be used to define the outer edges of the halo image (investigator adjusting based on subject feedback). Ascending and descending methods of limits will be used. This measurement takes about 10-15 minutes. Record values OD and OS, in mm (2 decimal places). Subjects will respond to a single-item post-halo questionnaire OD and OS: • How severe / intense was the halo that you experienced? Subjects will have the following response options: Severe, moderate, mild, not at all. |
| 4 | Repeat | The steps above will be repeated but with the alternate light source testing method. The investigator must allow at least 10 minutes to lapse before starting the second round of testing. |
| 5 | On-eye Light<br>Transmission | Measuring the in vivo light transmission (alternatively, the optical density) of ophthalmic lenses has been described in detail elsewhere using similar optical systems. The optical density (OD) of the test lens will be derived by comparing these threshold values to the rhodopsin curve, adjusted to a maximum OD equal to 0.35. This procedure obviously measures the density of all the ocular media. However, because the majority of the absorbance is due to the lens, the convention of referring to these values simply as lens density will be used. Given the extra time needed to perform this measurement, and the fact that on eye light transmission will be constant across all subjects (this reflects properties of the optical system and lenses, themselves, as opposed to visual performance of individuals wearing the lenses), these measurements will be taken in a small subset of subjects (n=5) who, when scheduled, report having enough extra time to complete the measurements. |

VISIT 2
Subjects must enter Visit 2 wearing their own contact lenses.

| | Visit 2: Treatment 2 | |
|---|---|---|
| Step | Procedure | Details |
| 2.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| 2.2. | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual correction in place. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 2.3. | Remove Habitual<br>Lens | If applicable, the subject's habitual contact lenses will be removed and stored in their own lens case. If they forgot to bring their lens case, one will be provided to them. |
| 2.4. | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If any of these slit lamp findings are grade 3 or higher, the subject may not continue at this time, but may return up to one additional time to determine eligibility. If discontinued a final examination must be completed. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 2.5. | Continuance after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. This refers to the concomitant medications and slit lamp biomicroscopy. If subject is deemed to be ineligible after two baseline attempts at Visit 2, proceed to Final Evaluation and complete all forms. |
| 2.6. | Lens Selection | Assign the study lens based on the randomization scheme. |

| Visit 2: Treatment 2 | | |
|---|---|---|
| Step | Procedure | Details |
| | | Select the contact lens power based on the refraction from Visit 1 or the final lens power from Visit 1. Record the test condition. |
| 2.7. | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Replace damaged lenses if applicable. |
| 2.8. | Lens Settling 1 | Allow the study lenses to settle at least 5 minutes before continuing. |
| 2.9. | Subjective Best<br>Sphere Over<br>Refraction | Perform subjective best sphere refraction over<br>the study lenses (adopt the maximum plus to<br>maximum visual acuity (MPMVA) approach. |
| 2.10. | Lens Power<br>Modification (if<br>applicable) | Adjust the lens power if the subject's best sphere over-refraction is not plano. For any power modification, repeat steps 2.7-2.9). One power modification is allowed. |
| 2.11. | Lens Settling 2 | Please wait for at least 10 minutes from final lens insertion to continue. |
| 2.12. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 2.13. | Visual acuity | Record the best corrected Snellen <u>distance</u> visual acuity to the nearest letter (OD and OS). Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 2.14. | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: • limbal exposure at primary gaze or with extreme eye movement • edge lift |

| Visit 2: Treatment 2 | | |
|---|---|---|
| Step | Procedure | Details |
| | | excessive movement in primary and up gaze insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up Note: if lens fit is unacceptable subject will be discontinued from the study. |
| 2.15. | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Visual acuity is 20/30 or better OD and OS 2. The lens fit is acceptable OD and OS 3. Investigator approval. If the Investigator does not approve the wearing of the study lenses for the psychophysical testing, then the study is terminated for that subject. |
| 2.16. | Lenses Worn in<br>Clinic | The lenses will be released for approximately two hours. 1. The subjects must wear both study lenses the entire time. 2. The lenses will be worn as daily wear only. 3. Rewetting drops are permitted if needed. Note: In the event a lens is lost or damaged, it will be replaced immediately. Note: A clinic-only-wear Patient Instruction Guide will be provided. |
| 2.17. | Sequence<br>Randomization | At Visit 2, all subjects will proceed to Psychophysical Testing B: This includes 2-point light threshold, haloes, and starbursts. Five subjects that are willing to undergo further in vivo light transmission testing will have this procedure performed. Following the psychometric testing by the co-investigator, the subject will return to the principal investigator to complete the study visit as described in steps 2.18 – 2.19. |

| | Visit 2: Treatment 2 | |
|---|---|---|
| Step | Procedure | Details |
| 2.18. | Lens Removal | The worn study lenses will be removed and discarded. |
| 2.19. | Exit Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. |
| | | Ocular adverse events shall be those that grade 3 or 4 on the FDA scale. The study monitored must be notified immediately. The AE will be followed to resolution. |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. |
| F.2 | Subjective<br>spherocylindrical<br>Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter and record the best corrected <u>distance</u> visual acuity to the nearest letter (OD, OS, and OU). |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pre-treatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit. |
| U.2 | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| U.3 | Entrance VA | Record the entrance distance visual acuity (OD, OS and OU) to the nearest letter. |
| U.4 | Subjective Sphero-<br>cylindrical<br>Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected <u>distance</u> visual acuity to the nearest letter (OD, OS, and OU). |
| U.5 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| U.6 | Exit Visual Acuity | Record the subject's exit distance visual acuity (OD, OS, and OU) to the nearest letter. |

### 7.4. Laboratory Procedures

The optical bench will be used to measure the light transmission characteristics for all worn Test lenses. The findings are for internal information only and will not be part of the final report.

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

Subjects are considered to have completed the study if they have completed all scheduled visits.

## 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol (e.g. Subject more than 2 days out of visit window).
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear (subjects missing more than 2 days of missed lens wear within a period 1 of week should be discontinued)
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject missed any scheduled study visits
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2. Collect all unused test article(s) from the subject.

Investigator will discuss with sponsor before enrolling any additional subjects if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: See section 3.3

Concomitant therapies that are disallowed include: See section 3.3

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

## 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)"
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site
- Lens replacements that occur due to drops/fall-outs
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)
- OD/OS indication, along with whether the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.

*Note 1* to entry: This definition includes events related to the investigational medical device or the comparator.

*Note 2* to entry: This definition includes events related to the procedures involved.

*Note 3* to entry: For users or other persons, this definition is restricted to events related to investigational medical devices." <sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

Serious Adverse Event (SAE) – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect
- Requires intervention to prevent permanent damage (the use of the test article resulting in a condition which requires medical or surgical intervention to preclude permanent impairment of the body structure or a body function). Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization

- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

*Note 1* to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

*Note 2* to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device." <sup>1</sup>

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

## 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 0)
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown
- Actions Taken none; temporarily discontinued; permanently discontinued; other

### 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge

### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of

severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities

## 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

#### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1. Reporting Adverse Events to Sponsor

#### **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

## **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

## 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

#### 13.5. Event of Special Interest

None

### 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation (SD), median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

## 14.2. Sample Size Justification

The plan is to enroll a maximum of 66 subjects with a minimum target of 60 subjects to complete. The sample size was chosen by the study responsible clinician and was not based on any empirical power calculation. Furthermore, a power calculation cannot be provided for any of the primary endpoints because no historical data is available. This data from this study will be utilized in the sample size calculations for any additional follow-up studies.

#### 14.3. Analysis Populations

### **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

### **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the per-protocol population set will be documented in a memo to file.

### **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

#### 14.4. Level of Statistical Significance

Each primary and secondary hypothesis will be tested individually using a type I error rate of 5%.

### 14.5. Primary Analysis

## <u>Light Scattering (Two-point Light Spread Function)</u>

This is defined as the minimum distance (mm) that two points of light are completely distinct. This threshold will be analyzed by a linear mixed model. Sequence of lens wear, lens type, age group, dominant eye and the interaction between lens type and age group will be included in the model as fixed effects. An appropriate covariance structure will be used to model the residual errors between measurements between eyes within a subject. The variance-covariance structure will be selected based on the finite-sample corrected Akaike's Information Criterion Corrected (AICC). The structure that returns the lowest AICC will be deemed the most appropriate structure. Covariance structures under consideration include:

- Unstructured (UN)
- Compound Symmetry (CS)
- Heterogeneous Compound Symmetry (CSH)

Heterogeneous covariance structures across lens type may be considered if necessary. The Kenward and Roger method (Kenward and Roger, 1997)<sup>15</sup> will be used for the denominator degrees of freedom.

Comparisons between lenses (Test inactivated vs Control and Test activated vs Control) will be carried out using 2-sided 95% confidence intervals constructed for the least-square mean (LSM) difference (Test – Control). Statistically significantly lower differences of the Test lens relative to the Control lens will be concluded if the upper limit of the 95% confidence interval is below 0. If the interaction between lens type and age is significant then comparisons between lenses will be made within age group.

#### Starburst

Starbursts will be quantified by the diameter of the light's lateral spread. A calibrated custom-made micrometer (two sides with reverse threading) will be used to spread two posts out from a central mid-point). Those posts can then be used to define the outer boundaries of the starburst image (i.e. the diameter). The diameter of the light's lateral spread will be analyzed and tested in the same manner as described for light scattering above.

#### Halos

<u>Halos will be quantified</u> by the diameter (mm) of outer edges of the halo image and is measured using the same micrometer as for starbursts and light scattering. The diameter will be analyzed using the same model as described for light scattering.

## 14.6. Secondary Analysis

#### Photostress Recovery Time (Seconds)

Photostress recovery time (PSRT) will be evaluated by exposing subjects to an intense light source (10-deg circular broad-band white at ~4.5 log Tds) and will be quantified as the time necessary to regain site of the grating after exposure.

PSRT will be analyzed using a linear mixed model. Sequence of lens wear, lens type, age group dominant eye and all the interaction between lens type and age group will be included as fixed

effects. An appropriate covariance structure will be used to model the residual errors between measurements between eyes within a subject. The variance-covariance structure will be selected based on the finite-sample corrected Akaike's Information Criterion Corrected (AICC). The structure that returns the lowest AICC will be deemed the most appropriate structure. Covariance structures under consideration include:

- Unstructured (UN)
- Compound Symmetry (CS)
- Heterogeneous Compound Symmetry (CSH)

Heterogeneous covariance structures across lens type may be considered if necessary. The Kenward and Roger method (Kenward and Roger, 1997)<sup>15</sup> will be used for the denominator degrees of freedom.

Comparisons between lenses will be carried out using 2-sided 95% confidence intervals constructed for the least-square mean (LSM) difference (Test – Control). Statistically significantly lower differences of the Test lens relative to the Control lens will be concluded if the upper limit of the 95% confidence interval is below 0. If the interaction between lens type and age is significant then comparisons between lenses will be made within age group.

### Disability Glare Threshold (Change in log relative energy level)

Glare disability threshold (GDT) (change in log relative energy level) will be evaluated by exposing subjects to various intensity of a white-light annulus (10-geg diameter) and will be quantified by the log relative energy level necessary to obscure a central target.

GDT will be analyzed and tested in the same manner as described for PSRT.

#### Discomfort Glare (change in palpebral fissure height (mm))

Glare discomfort (GD) will be evaluated by squint response of the extraocular muscles and by a subjective questionnaire regarding the patients' comfort. Squint response will be captured by using a high-resolution camera for each subject eye. The resultant videos will then be analyzed as still frames. Squint response will be quantified as the calculated ratio of the height of the palpebral fissure under normal light conditions compared to maximal squint produced during the Photostress exposure. GD will be analyzed in the same manner as described for PSRT.

Comparisons between lenses will be carried out using 2-sided 95% confidence intervals constructed for the least-square mean (LSM) difference (Test – Control). Statistically significantly higher differences of the Test lens relative to the Control lens will be concluded if the lower limit of the 95% confidence interval is above 0. If the interaction between lens type and age is significant then comparisons between lenses will be made within age group.

#### Heterochromatic Contrast Threshold (HCT)

Heterochromatic contrast thresholds will be evaluated using a variable wavelength central target presented on a short-wave (460nm) sky-light background and will be quantified by the amount of light absorbed by the macular.

HCT will be analyzed and tested in the same manner as GD.

## 14.7. Other Exploratory Analyses

In vivo light transmission and slit lamp findings will be descriptively summarized for each lens type.

### 14.8. Interim Analysis

There will not be an interim analysis conducted on this study.

## 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 10 imputations.

#### 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

#### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

The follow data testing/measurements will be calculated and entered into the EDC at the study site.

- Light Scattering
- Starburst
- Halos
- Photostress Recovery Time
- Disability Glare Threshold
- Discomfort Glare
- Heterochromatic Contrast Threshold

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011. 1

#### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the

clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

## 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

## 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies

- Clarifying questions regarding the study
- Resolving study issues or problems that may arise
- Reviewing of study records and source documentation verification in accordance with the monitoring plan

#### 18. ETHICAL AND REGULATORY ASPECTS

## 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

## 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

## 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

### 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

#### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA)<sup>19</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution
- Case Report Form signature
- Completion of any follow-up action items

#### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 22. REFERENCES

- ISO 14155:2011: Clinical investigation of medical devices for human subjects Good clinical practice.
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP): http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. http://www.wma.net/en/30publications/10policies/b3/index.html.
- 4. United States (US) Code of Federal Regulations (CFR). In <a href="https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR">https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR</a> (Ed.).
- Renzi-Hammond, L.M. and B.R. Hammond, The effects of photochromic lenses on visual performance. Clinical and Experimental Optometry, 2016. 99(6): p. 568-574.
- 6. Artal, P. and R. Navarro, *Simultaneous measurement of two-point-spread functions at different locations across the human fovea*. Applied Optics, 1992. **31**(19): p. 3646.
- 7. Avant, L., Vision in the Ganzfeld. Psychological Bulletin, 1965. **64**(4): p. 246-258.
- 8. Ritschel, T., et al., *Temporal Glare: Real-Time Dynamic Simulation of the Scattering in the Human Eye.* Computer Graphics Forum, 2009. **28**(2): p. 183-192.
- 9. Buch, J. Clinical Study Protocol Evaluation of Lenses Made with new UV-Blocker 2018 09 January
- 11. Franklin, R. Clinical Study Report Proceedings of Temporally Asymmetric Interocular Blur. 2017 04 January
- 12. Sayre, R., et al., *Spectral comparison of solar simulators and sunlight.* Photodermatol Photoimmunol Photomed, 1990. 7: p. 159-165.
- Mecherikunnel, A.T. and J.C. Richmond. (1980). Spectral distribution of solar radiation. Greenbelt, Maryland.
- 14. Hammond, B., et al., Contralateral comparison of blue-filtering and non-blue-filtering intraocular lenses: glare disability, heterochromatic contrast, and photostress recovery. Clinical Ophthalmology, 2010: p. 1465.
- 15. Sheedy, J.E., et al., *Is all Asthenopia the Same?* Optometry and Vision Science, 2003. **80**(11): p. 732-739.

- 16. Stringham, J.M., K.J. O'Brien, and N.T. Stringham, *Macular carotenoid* supplementation improves disability glare performance and dynamics of photostress recovery. Eye and Vision, 2016. **3**(1).
- 17. Nahar, N.K., et al., *Objective Measurements of Lower-Level Visual Stress*. Optometry and Vision Science, 2007. **84**(7): p. 620-629.
- 18. Gowrisankaran, S., J.E. Sheedy, and J.R. Hayes, *Eyelid Squint Response to Asthenopia-Inducing Conditions*. Optometry and Vision Science, 2007. **84**(7): p. 611-619.
- 19. Health Information Portability and Accountability Act (HIPAA). In https://www.hhs.gov/hipaa/for-professionals/privacy/index.html (Ed.).
# APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)





2

| Protocol 6100 | Johnson & Johnson Vision Care, Inc. | Confidential |
|---------------|-------------------------------------|--------------|

3



# **APPENDIX B: PATIENT INSTRUCTION GUIDE**

The Patient Instruction Guide will be provided separately.

# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

• Acuvue OASYS Brand Contact Lenses

If vision is acceptable, perform a sit tamp-examination to assess adequate fit (sentration and movemen ). If it is acceptable, disperse the lesses instructing the patient to return in one seek for examesoment, tipes dispersing and follow-up information in PATIENT MANAGENERNI).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are wallable for download at

### TORIC FITTING GUIDELINES

A though most aspects of the fitting procedure are identical for all types of soft contact lenses; including torics, there are some additional steps and/or rules to follow to assure the properfit of toric lenses.

The onlynew steps you must follow in prescribing AGUALE CASYS\* for ASTIG-MATEM contact lenses are that you must determine the stability repeatability are drift angle of the lens axis so that you can prescribe the correct lens axis (or your

1. Localethe Orientation Marios.
To help distarmine the proper orientation of the toric lens, you'll find two primary to very occurrent the proper of entation of the folial feet by \$0.00 ft and \$0.00 f

Vifigure 1

Volumed a bornioroscope and a 1 mm or 2 mm para leiepped beamto highlight the maries when the lives is titled to the eye. There are a number of a contribute you can be not prove the visible of the 5 circle instance, and a contribute you color beam and medium magnification 100x or 150, slowly goan down the law, looking state leien the devict furnishment at the action laminated area. Backlighting the mark this way should make it more visible. Some times a manipulating the lower if demands are considered in the contributed area.

2. Observe Lens Rotation and Stability Observe the position and stability of the "boltom" mark, it usually stabilizes at

the 6 of dock position. If it does, calculation of the lens power will be straightforward. The 6 of dock position is not a "must"; however, the absolute requirement is that the axis position be stable and repeatable. A low the lenses to settle for about 20 minutes with the correct power is

Alow the investio satisface about 20 minutes with this correct proved enters in place. What scropes he received produced to the particul root stupp. Assess the particul root stupp. Assess the particul root stupp. Assess the particul root stupped as a particul root stuffer investigation of the satisface and particul root stuffer produced as particul root stuffer investigation. Then have the nat and distance objects, observe the reactions. Only within these vision tests or completed mobile the particul root students of read particular the particular reactions to grape price (e.g., 1) powerfron copyl at first and then graduate to nesign that finally private types as the

A fer the patient's performance under the above conditions is completed, it of visual souty and reading ability under conditions of moderately dimillum

An initial untworable response in the office, while indicative of a guarded prog-nosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

4. Adaptation
Visually demanding situations should be assolided during the initial wearing period. A patient may at first experience are middle turned stoon, dischess, has able as one as and a feeting of slight three sistence. You should explain the adaptation all symptoms to the patient. These symptoms may last for a brief minute or for award seeks. The longer these symptoms preside, the power the prognosis. for successful a displation

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable familiar environment such as in the home.

Some patients feel that automobile driving performance may not be op imal during the adaptation process. This is particularly true when driving at night. Before driving, a motor veried, at truty per recommended that the patient be a passenger first to make sure that the vision is satisfactory for operating an a comobile. During the first several weeked of ware pith or adaptation is occurring the combined of the patients of the It may be advisable for the patient to only drive during optimal driving condi-tions. After adaptation and success with these activities, the patient should liable to drive under other conditions with caution.

### D. Other Suggestions

The success of the monovision technique may be further improved by having the passent follow the suggestions below:

. Have a third contact lens (distance power) to use when critical distance viewing

Have a third contact lens (near power) to use when critical near viewing is needed.

2. Chemonth post-dispensing

The mark may stablibe some what left or right (\$int) of the vertical meridian and all enable you to iff a loric tens for that eye, as long as the tens always returns to the same "drift axis" position after setting. The deviation can be compensale difor in the final prescription. Your objective is to ensure that whatever position the initial lens assumes near 6 of clock, this position must be stabland repositable. With full ever povement or heavy bink, you may see the n swing away, but they must return quickly to the original stable position. If the lens does not return quickly, you may need to select a different lens.

### Assessing Rotation

Integrating recursion in the page 32 and old dail and eway hour represents a 30° interval. If the orientation mark of the initial interstablibles comments, list or right of the vertical position, the first list set of end of the list was devicted in . You can use an action of olde in the set flamp or uses an exception of the first in a special of tall fame to measure or a district the "office and of the set of the

To compensate for this "drift", measure or estimate the "drift", then adid or subtract it from the refis cities axis to determine the correct cylinder axis. Use the LARS Left Add. Right Subtract) method to determine which direction to

### B. How to Determine the Final Lens Power

When the diagnostic lens has its axis signed in the same meridian as the patient's refractive axis, a sphero cylindric all over-refraction may be performed and visual acually determined. However, in the case of crossed axes, such as arts values about 9 describer for critical value in the Case or critical about 9 describer in which the diagnostic lens add in it of Sent from the pulser for reflective adds, it is not additionable to over-reflect because of the difficulty in computing the results of power in this power in the power in the power in the sphere. In the opinion, the counterrapty one presents defined up to ever in the sphere. In the opinion of the present is as the counterrapty one presents as the counterrapty of durating to the patient, as of its more practical value of presents as servation by the day to power in the presents as servation by the day to power in the presents as the counterpart of the patients. So, here is how to determine the final lens power

### For the Cylinder:

Adjust the axis by the drift angle using LARS. Choose a cylinder that is  $\le 0.25D$  from the refractive cylinder.

### Example 1

C.S. -2.00 - 1.00 x 180 20/20

for specific visual basics may improve the success of monovision correction.

This is particularly applicable for those patents who cannot pass state drivers licensing requirements with monovision correction.

. Make use of proper illumination when carrying out visual basics.

Monovision fitting success can be improved by the following suggestions: Revenue the distance and near eyes if a patient is having to uble adapting.
 Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for preabyopic patients.

. Emphasize the benefits of clear near vision and straight ahead and upward gaze with monovision.

he decision to fit apatient with a monovision correction is most appropriately left the Eye Care Professional in conjunction with the patient after carefully consider

# All patients should be supplied with a copy of the PAT ENT INSTRUC-TION GUIDE for these lenses. Copies are available for download at www.

### PATIENT MANAGEMENT

PROVIDE THE PATIENT WITH A COPY OF THE PATIENT INSTRUCTION QUIDE FOR THESE LENGES. REMENTHESE INSTRUCTIONS WITH THE INTENTSO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBE WEARING AND REPLACEMENT SCHEDULE (DISPOSABLE OR FREQUENT REPLACEMENT).

Recommend an appropriate cleaning and dain/ecting system and provide patient, with instructions requiring proper lens care. Chemical or hydroge percode dishrection is recommended.

### Follow-up Examinations

Follow-up care thesessary to ensure continued successful contact lens weary should include notifice periodic progress examinations, management of specific problems; framy, and a review with the patient of the wear schedule, lens replacement, schedule, and proper lens case and handing procedures.

Recommended Follow-up Examination Schedule (complications and specific problems should be managed on an individual patient basis):

One week from the initial lens dispensing to patient

it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, sucheck until stable. Gheck the orientation of the axis mark. If the bottom axis mark is in the 6 of clock position on both eyes, choose the appropriate cylinder ax listed previously. If the lens has not yet stabilized, neche ckuntil stable. Here is the PorPres

OD. -2.50 -1.25 x 180 OS. -2.00 -0.75 x 180

### Example 2

Co. — 1.10 - 1.00 / 1.0 The fitting indicates the following:

Right Eye:
Gompensale the 10" axis drift by adding it to the manifest refraction axis.
Have in the for exemplant -3.00 -0.75 x 100

Left Eye
The lens on the left eyes in own good centration, movement and a consistent tendency for the mark to drift right by 10° from the 6 o'd coic position. wing aforced blink. Singethe manifest refraction as led for a power of -4.750, a djust for the vertex distance and reduce the sphere by 0.25 D and prescribe the -1.750 cylinder. Compensate for the 10° axis drift by subtacing it from the manifest refraction.

Here is the Rx Prescribed:

OS -450-175 v 80 If vision is acceptable, performs sit i amp examination to assess adequate fit contration and movement). If it is acceptable, dispense the lenses instructing the pale int to return in one weekfor reassessment (see a dispensing and follow up information in PATENT MANAGEMENT).

# All patients should be supplied with a copy of the PATIENT INSTRUCTION OU DE for these lenses. Copies are available for download at

NOTE: More frequent or additional follow-up visits may be recommended for patients on an extended was schedule. Preferably, at the follow-up visits, lenses should be worm for at least sich our.

If the lenses are being worm for continuous weat the ecomination should be performed as easy as possible on its emorning following overnight weat.

commen ded Pro cedures for Follow-Up Vist: 1. So icit and record patient's symptoms, if any.

We saw visual soully monocularly and bin ocularly at, distance and near with the contact lesses. Performan over-extraction at distance and near to check for residual extractive error.

With the biomicroscope, judge the lens fi ting chass deristics (as described in the GENERAL FITTING GUIDELINES) and evaluate the lens surface for deposits and damage.

Following lens removal, examine the comes and conjunctive with the biomi-coscope and fluorescein (unless contraindicated). The presence of vertical corneal strise in the posterior central corneal and/ or corneal necessicalization is in dicative of excessive corneal edema. \*The presence of comesi staining and/or imbal-conjunctival hyperemia.
can be indicative of an unclean lens, a reaction to solution presentatives

velens wear, and/or a poorly fitting lens. Papillary conjunctival change a may be indicative of an unclean and/or

Periodically perform liverate metry and aplectacle refractions. The values should be recorded and compared to the baseline measurements.

If any observations are almormal, use professional judgment to allevials the problem and restore the eye to optimal conditions. If the orbina for surceast lift are not attained during any follow-up examinations, repeat the patient's trial fitting procedure and refit the patient.

### WEARING SCHEDULE

The wearing and replacement schedules should be determined by the Eye Gae Professional Regular checkups, as determined by the Eye Gae Professional, ar

### For Daily Wear:

or busy reser. Taken's ten't to overwest the lenses in it sily. The Eye Care Professional should mehasise the importance of adhering to the initial maximum we aring schedule, bushmum wearing it me should be defermined by the Eye Care Professional base pon it he palletts; physiological eye condition, because in dividual wap ores to

### MULTIFOCAL FITTING GUIDELINES

Multifocal contact, larses may produce compromise to Valon under certain ole umatanose and the patient should understand in at they might not find the valors acceptable in specific situations (a.e., reading a menu in a dire in statusard driving at night in rainyly loggy conditions (e.e.). The webs, caution should be asked as delent he patient in sealing the correction for the first that of all causes and the specific situations. e and can derive may passent is sweating the correction of the instruction and they are familiar with the vision provided in invisually for basinging environments. Goographical and servironmental visual demands should be considered. If they patient is quites or tribuil a business of their individual is a should be desired. If they patient is quites or tribuil a business of their individual in the patient can function adequately with the ACUIVLE CASIFS\* for PRESENTIAR contract claims. When may not be optimal for activities such as:

visually demanding situations auch as operating potentially dan genous machinery or performing other potentially hazardious activities; and

me, executorists (e.g., driving at night). Patients who cannot pass their state driver's loanse requirements with these lenses should be adulted to not drive with this correction. CR may require that adultional over-correction be prescribed. 2. driving sutomobiles (e.g., driving at night). Patents who cannot pass their

These lenses are not recommended for patients who have -1 000 or greater of refractive cylinder as this level of uncorrected cylinder may lead to additional compromise.

These lenses are available in the following ADD powers:

\* Lens "LON" = "low" ne ar ADD len s (Max +1.25 ADD)

\* Lens "WID" = "medium" near ADD lens (Max +1.75 ADD) \* Lens "HGH" = "high" near ADD lens (Max+2.50 ADD)

### B. Pitting Instructions

1. Determine the following: Eye domin ance (the metho do described in MCNOVISION FITTING QUID E-LINES may be used)

### + New ADD 2. Select the initial trial lens as follows:

The maximum suggested wearing time for these lenses is:

| DAY | HOURS |
|-------------|------------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | a I waking hours |

# t is recommended that the contact lens wearer first be evaluated on a daily wear

schedule. If successful, then a gradual introduction of extended wear can be followed as determined by the prescribing Eye Gare Professional. These lenses have been approved for extended wear up to 6 nights/7 days of continuous wear. Not all patients can achieve the maximum wear time.

For Therap-suite ien's wear, close supervision by the Eye Care Professional in necessary. These ien see can be worn for extended wear for up to 6 nights/7 of continuous wear. The Eye Care Professional should determine the appropri wearing time and provide specific instructions to the patient regarding lens care,

### REPLACEMENT SCHEDULE

When prescribed for daily wear (frequent replacement), it is recommende lenses be discarded and replaced with a new lens every? weeks. Howe Care Professional is en couraged to determine an appropriate replacement based upon the wapportee of the patient.

When prescribed for dispossible wear, the replacement schedule should be determined by the Eye Gase Professional based upon the patients history and their coular examination, as well as the practitioner's experience and cinical judgment. Once removed, it is secommended that the lens semain out of the eye for a period of set of overnight, or longer and be discarded in accordance with the prescribed. wearing schedule. The Eye Care Professional should examin eithe patient during the early stages of extended wear.

ADD: +0.75 to +1.25 use a "LOW" near ADD lens on each eye ADD: +1.50 to +1.75 use a "MID" near ADD lens on each eye ADD: +2.00 to +2.50 use a "HQH" near ADD lens on each eve

3 Allow the lens to settle for a minimum 10 minutes. 4. Assess distance and near vision bin ocularly and monocularly.

 Demonstrate the vision under various lighting conditions (normal and decreased illumination) and at distance, intermediate and near. Make adjustments in power as necessary (see Mutificial Troubleshooting below). The use of han diheld trial lenses is recommended.

 If distance and near-vision are acceptable, perform a sit tamp examination to assess adequate it (sentration and movement). If it is acceptable, dispense the lanses instructing the patient to return in one week for reassessment, (see dispensing and follow-up information in PATIENT MANAGEMENT).

Unacceptable Near Vision:
Determine the amount of additional plus, or less minus, over one or both eyes
that is acceptable, while checking the effect on distance and near vision. If
vision is all not acceptable, change the non-dominant eye to the next highest.
ADDI present

Unacceptable Distance Vision: Determine the amount of additional minus, or less plus, over one or both eyes

Determine the amount or adaptions mustic, or easily and, over one or force that it is acceptable while checking the effect on distance and near vision. If vision is still not acceptable, change the dominant eye to the next lowest A. power. If the patient is searing two low ADD lenses, change the dominant eye to a sphee lens with a power equal to the spherical equivalent distance ye

prescriptor. Distance and New Yislan: Determine the amount of salidonal plus and or minus over one or both eyes to be amount of salidonal plus and or minus over one or both eyes that is acceptable which done high exide con distance and near vision. If salidonal plus and/or minus is not required, change the less power in the dominant eye to the next (accept ACD power and the less power in the non-dominant, eye to the next high-set ACID power, if app isable.

Al patients should be supplied with a copy of the PATIENT INSTRUCTION GUID E for these lenses. Copies are available for download at

### LENS CARE DIRECTIONS

Nhan lenses are dispersed, the Eye Care Professional should provide the patient, with appropriate and a dequate warmings and instructions in accordance with the neighbours of the terminal stress of the second second second second should recommend an appropriate can system talowel to the patient's individual

For complete in 6 must on concerning contact lens handing, care, cleaning, dish-fecting and storage, wifer to the Patient Instruction Guide for these lenses. Copie we contain to the deservation of a season extracts. com

### For Lens as Prescriped for FrequentReplacement Wear

The Eye Care Professional should seview with the patient, lens care directors is clearing, disinfecting and storing, including both basic clears care information an specific instructions on the lens care regimen recommended for the patient. For Lens as Prescribed for Disposable Wear:

### The Eye Gare Professional should review with patients that no cleaning or disinfecton is needed with disposable lenses. Patients should always dispose of lense when they are removed and have replacement lenses or speciacles are label. Lenses should only be cleaned in set and districted on an emergency basis. when replacement lenses or spectacles are not available

Gare for a Dried Out (Dehydrated) Lens If the frequent, replacement, lens is off the eye and exposed to air from 90 minutes to 1 hour or more, its surface will become day and gladius lybecome non-welfing. If this should occur, discard the lens and uses new one.

### Gare for Sticking (Non-Moving) Lenses

were or accounting two-menting Lanses. With the size of the paper is should be instructed to apply a few drops of the recommended luteriating or review ting solution directly to the seed or representation of the size begins to move fewly on the eye before a moving it in one movement of the land continues after a few minutes, the patent should immediately contact the fig. Care in Professional.

### EMERGENCIES

gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the pa-fent should: FLUSH EMES INVECIDATELY WITH TOP WOUTH AND INVECTIVELY CONTACT THE EME CAME PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY ROOMS WITHOUT DRIVE.

### MONOVISION FITTING GUIDELINES

### A. Patient Selection

Monovision Needs Assessmen For a good provise, the publish, should have a dequately come ded distance and near visual acuty in each eye. The amblyopic pastent or the pastent with significant astigmast m (greater than 1.000) in one eye may not be a good candidate for monovision correction with these learness.

Coupational and environmental visual demands should be considered. If the patient requires critical vision frieural sculty and stereopsist, it should be determined by that whether this patient, can fun of on adequately with monoul sion correction. Monovision contact in ma wear may not be optimal for activities such

driving sullo mobiles (e.g., driving at nigh). Patients who cannot pass their state driver's loanse requirements with monovision correctionshould be advised to not drive with this correction, CR may require that additional over-correction be prescribed.

Particular Biological Properties of the Control of with the vessor provised in vessally challenging environments (e.g., was dreg a menu in a dimensionaria, ching at right in rainyloggy conditions, etc.). During the fitting so-cess, it is no essessy for the patient to realize the disad-varianges are well as the advantage so-of-dear new vision and straight ahe ad-upward gaze that monovision contact linears provide.

### B. Eye Selection

1. Ocular Preference Determination Methods Method 1: Determine which eye is the "sighting eye." Have the pastent point to an object at the far end of the aroom. Governmence. If the patient is still pointing directly at the object, the eye being used is the dominant pighting) eye.

### HOW SUPPLIED

\* ACUVUE OA SYS\*: base ourve, power, diameter, lot number, and expl

· ACLIVUE OA SYS\* for A STIGMATISM: base curve, power, diameter

· ACUVUE OA SYS\* for PRESBYOPIA: base curve, power diameter ADD.

### REPORTING OF ADVERSE REACTIONS

All serious adverse experiences and adverse reactions observed in patients was ing these lenses or experienced with the lenses should be reported to

Johnson & Johnson Vision Gare, Inc.



In Canada: Johnson & Johnson Vision Care, division of Johnson & Johnson, In LISA: Johnson & Johnson Vision Care, In

AGUVUE CASYS\* and HYDRAGLEAR\* are trademarks of Johnson & Johnson Vision Care Companies.

Method 2: Determin ewhich eye will accept the added prover with the least reduction in vision. Place a hand-hald that lens equal to the specified near ADDI from of one eye and then the other whells the distance will not one eye and then the other whells Determine wealther the pudent fundoms best with the near ADDI lens over the right of this dyna.

Other methods include the refractive error method and the visual demands

2. Refractive Error Method:
For anisometropic correction, it is generally best to fit the more hyperopic (ess:
myopic) eye for distance and the more myopic (less: hyperopic) eye for near.

 Visual Demands Method
 Consider the patient's occupation during the eye selection process to determine the offical vision requirements. If a patient's gaze for near tasks is usus ly none direction, correct the eye on that side for near.

# <u>Framelie:</u> A secretary who places copy to the left side of the dask will function best with the near lens on the left eye.

### C. Special Fitting Characteristics

Unlibbrasi Lens Cornection
 There are circumstances where only one contact lens is required. As an excample, an errorator pic patient would only require a near lens while a bit also at mycope may only require a distance lens.

Example: A presisyopic emmetropic platent who requires a +1 75D ADD would have a +1.75Diams on the rear eye and the other eye left without a lens. A prestyppic patient requiring a +1.50D AXD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.

2. Near ADD Determination.
Aways prescribe the lens power for the near eye that provides optimal near
acuty at the miscoint of the patent's habitual reading distance. However, when
more its area of the patent's habitual reading performance, prescribe the
least plus great missage of the power.

### 3. Thial Lens Fitting A trial fiting is performed in the office to allow the patient to

ction. Lenses are fit a coording to the GENETIAL RITING CLIDELINES for base curve selection in this Package Insert.

Case history and standard dinical evaluation procedure should be used to distamine the prognosis. Date mine the distance correction and the near correction. Next determine the near ADD. With trial larges of the proper power in place, do serve the reaction to this mode of correction.

IMPORTANT: Pleme read carefully and keen this

This Package Insert and Fitting Gu de is intended for the Eye Care Professional, but should be made available to patients upon request.

The Fire Care Professional should provide the natient with the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at www.acuvue.com.



BRAND CONTACT LENSES ACUVUE OASYS+ Brand Contact Lenses ACUVUE QASYS® Brand Contact Lenses for ASTIGMATISM

ACUVUE QASYS\* Brand Contact Lenses for PRESBYOPIA nofilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker for Daily and Extended Wear GAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner.

JJVC CONFIDENTIAL CR-6100, v 2.0 Page 80 of 117

The following symbols may appear on the label or carton

| SYMBOL | DEFINITION |
|---|---|
| (II)A | Consult Instructions for Use |
| - | Manufactured by or in |
| 쎈 | Date of Manufacture |
| <u> </u> | Use By Date (expiration date) |
| LOT | Batch Code |
| ET LE | Sterle Using Steam or Dry Heat |
| DIA | Diameter |
| BÇ | Base Curve |
| В | Diopier (ens power) |
| CYL | Cylinder |
| AXES | Aoás |
| MAX ADD | Near ADD |
| LOW | "Low" Near ADD |
| MB | "Medium" NearADD |
| нан | "High" Near ADD |
| 2004 | Quality System Certification Symbol |
| Ç. | UV-Blocking |
| 0 | Fee Paid for Waste Management |
| R <sub>C</sub> ea | CAUTION: U.S. Federal law restricts this device to<br>sale by or on the order of a licensed practitioner |
| 2 | Lens Crientation Correct |
| Ă | Lens Crientation Incorrect (Lens Inside Out) |

### Disc and Date on Multi-Purpose Solution Bottle Instructions for Use

- The Disc ad Daterefers to the time that the patient can safely use contact, lens care product after the bottle has been opened. It is not the same as the expiration date, which is the last date that the product is still effective before
- WARN NO:

- o avoid contamination, DC NOT to uch tip of container to any surface. epiace cap after usin g.

### Instructions for Use

WARN NO-

- Rub and rince lenses for the ecommended amount of time to help prevent
- Never use water, sains solution, or reweiting dilops to disinfect the lenses. These solutions will not disinfect the lenses. Not using the ecommended disinfectant can lead to severe infection, vision loss, or bindhess.

### · Lens Case Care

- drame only accusion accordant, with dealer, Revenue is stated. Ceasing an be afollowed by inning with feath, sairel addistributing solutions (review use water) and wiping the term cases with feath, clean tissue is recommended. Never air dry or recap the lens case lifes after use without any additional cleaning methods. If air drying, be sure that, no residual solution remains the cleaning methods. If air drying, be sure that, no residual solution remains the cleaning methods. If air drying, the sure that, no residual solution remains the cleaning methods. If air drying, the sure that, no residual solution remains the cleaning methods are supplied to the cleaning that the cleaning dearing methods. If air drying, be sure that, no residual so lution remains in the case before allowing it to air dry. Replace the lens case according to the directions provided by the Eye Gase Professional or the manufacturer's labeling that, accompanies the case.

AGUNUE CASYS\* Brand Contact Lenses; the AGUNUE CASYS\* Brand Con Lenses for AST GMAT SM, and the AGUNUE CASYS\* Brand Contact Lenses oct Lenses for AST Geven gav, an or PRESBYCPIA are soft (hydrop) or multi focal lemses and include HYDEVICIENT PLUS Technology. The lemses are assumed in the deliverse and include HYDEVICIENT PLUS Technology. The lemses are made of a claim on hydrogol material containing an internal wetting agent with visibility tinted UV absorbing monomer.

These lenses a etinted bias using Residive Blue Dye #4 to make the lenses mole visible for handing. A bercotriscol eUV absorbing monomer is used to block UV

| a Properties: | |
|--------------------------------|-------------|
| Specific Gravity (calculated): | 0.98 - 1.12 |
| Rehactive Index | 1.42 |
| Light Transmitance: | 85% minimum |
| Surface Character: | Hydrophilic |
| Water Gontent: | 38% |
| Oncore Burecohillo | |

103 x 10<sup>11</sup> (sm²/sed) (ml O/ml xmmHg) @ 15°G Fattibiounds y corrected, edge corrected) Fatt (bounds y corrected, no n-edge our enterth 122 x 10 <sup>(1)</sup> (cm²/sec) (mi O /mi xmmHg) @ 35 °G

12.0 mm to 15.0 mm

varies with power

### Lens Parameters: Diameter Range:

 Genter Thickness: Spherical Power Range

7.85 mm to 10 00 mm Daily Wear: -20.00 D to +20.00D Extended Wear: -20,000 to +14,000 Multifo cal ADD Power Range: +0.25D to +4.00D -0.25D to -10.00D

 OyinderPowerRange: Axis Range:

Do not sto element or rime lens cases with water or any non-sterile solution. Only finish multi-purp cos solution should be used to prevent contamination of the lenses or lens case. Use of non-sterile solution can lead to severe infective.

### PRECAUTIONS

Special Precautions for Eve Care Professionato

- Due to the small number of patients enrolled in clinical investig at on of lens es, all refra dive powers, design configurations, or lens pla ameters availab in the lens material are not wall usted in significant numbers. Consequently in the serial majerial are not eaclused in agreement, numbers. Lo majerial when selecting an apper prisid send design and pas mellers, the Eye Care Profe solonal should consider all characte takes of the lens that can affect lens performance and coulder health, including copy any permeability, welltak ty, central and periphe all thickness, and optic zone diameter.
- The potential impact of these factors on the patient's ocale health hould be carefully weighed against the pallent's need for whactive on ector; therefor e, the continuing ocale health of the pallent and less performance on the eyesth ould be carefully monitored by the ple sorbing Eye Care. Producing the carefully monitored by the ple sorbing Eye Care.
- Patient's who wear these lenses to correct pleabyopis using monovision may not achieve the best corrected vious as utility for either fair or near siston. Visual equinments vary with he hiddidata and should be comisitered when selecting the most appropriate type of lens for each patient. Flu crescein, a vellow dive, should not be used while the lenses are on
- the eyes. The lenses absorb this dije and become discolored. Whenever fluorescen is used in eyes, the eyes should be flushed with a sterile saline solution that is recommended for in-eye use.
- Eye Care Professionals should inst, uct the patient to remove lenses immediately if the eyes become red or initialed.

### onals should carefully instruct patients about the followare regimen and a slety precaution

- . Before leaving the Eve Core P ofession of soffice, the patient should be able to promptly remove the lenses or should have someone else available who can remove the lenses for him or her.
- . DO NOT use if the sterile blister package is opened or damage di
- Always wash and rinse hands below handling lenses. Dion of get oss lotions, scaps, cleams, deciderants, or sprays in the eyes or on the le

### AVAILABLE LENS PARAMETERS

The ACUNUE CASYS\* Brand Contact Lenses are hemispherical shells of the

following dimensions: Genter Thickness: Minus Lens - varies with power (e.g. -4.000: 0.070 mm)
Plus Lens - varies with power (e.g. +4.000: 0.168 mm) 8.4 mm 8.8 mm -0.50D to -6.00D (n 0.25D

-6.50D to -12.00D (in 0.50D +0.50D to +6.00D in 0.25D The AGUVUE CASYS\* Brand Contact Lenses for AST QMATISM are hemitoric shells of the following dimensions:

Center Thickness: Minus Lens , varies with power is a .4 000: 0.000 month Plus Lens - varies with power (e.g. +4.000: 0.172 mm

+6.500 to +8.000 in 0.500 incremental

plane to -6.00D (in 0.25D increments) -6.50D to -9.00D (in 0.50D increments +0.25D to +6.00D in 0.25D increment: Ovinder: -0.75 D. -1.25 D. -1.75 D. -2.25 D. -2.75 D Axis: 10" to 180" (in 10" in crements)

The ACUIVUE CASYS\* Brand Contact Lenses for PRESBYCPIA are he

### 14.3 mm

Center Thickness: Minus Lens - varies with power (e.g. -4.00D: 0.070 mm) Plus Lens - wries with power (e.g., +4,000): 0,168 mm) BaseCurve 8.4 mm

-9.00D to +6.00D (in 0.25D in coments) +1.25 LOM: +1.75 (MDI: +2.50 HGH)

### is best to put on lenses befoe putting on makeup. Water-based cosmetics are less likely to damage lenses than oil-based products.

- DC NOT touch contact lenses with the fingers or hands if the hands are not fee of fo eign materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.

- Never use tweezers or other tools to serious lenses from the lens container unless specifically in dicated for that, use. Side the lens up the side of the sow until it, is free of the container.
- Do not touch the lens with fingernalis.
- Close supervision is necessary for the Therapeutic use of these lenses.
   Coute medications used during t eatment with a bandage term should be closely monitored by the Eye Clase Poisson at No ordan out are conditionary to Be Eye Clare Prolescion at Will lines to and remove the lenses. In these cases, patients a hold be instructed not to handle the lenses thereally a terminate and the conditional conditions.

- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Gare for Sipking (Non-Moving) Lenses". The lens should move feely on the eye for the continue directly of the eye. If non-movement, of the lens continues, the patient should be instructed to immediately consult his
- Never wear lenses beyon dith a period recommended by the Eye Gare The patient, should be a divised to never allow anyone else to wear the enses. They have been prescribed to fit their eyes and to correct their vision to the dieg elenecessary. Shis inglances gleatly increases theich ance of eye
- If sercool products, such as hair spray, are used while was inglences, exercise caution and losep eyes closed until the spray has settled.
- Avoid all harmful or initiating vapo is and furnes while we aring lenses
- Different solutions cannot always be used to gether and not all solutions are safe for use with all lenses. Use only recommended solutions.
- . Chemical disinfection solutions should not be used with heat unless

### TRANSMITTANCE CURVE



WARTLENGTH beaningted neifform measurems a takenthrough the certail \$5 mm portion or the trianed Olera. 6.05 mm center thistorium.

 Lemman, S., Raudant Energy and the Eye, Machillan, New York, 1980, p. 58, Space 3:31
 Wilster, M., Hitchina, VM., Optical Radiation and Valual Health, CR CP ess. Space Ration, Rollida. WARNING: UV absorbing contactionses are NOT substitutes for pro tive UV absorbing eyewear, such as UV absorbing goggles or sungla

because they do not completely cover the eye and surro

### patient should continue to use UV also orbing eyewear as directed. ACTIONS

The transmittance chis acteristics are less than 1 % in the UVB range of 280 nm to 3 to nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire

NOTE: Long-term exposure to UV radiation is one of the risk factor GITEL Long-term expeciative to LIV radiation is one of the risk factors is socialed with cataracta. Exposure in based on a number of factors ich as environmental conditions (altitude, geography, cloud cow et and enonal factors (alternal and nature of outdo or activities). LIV radiation intact lenses help provide protection against harmful LIV radiation.

- . Do not change solution without consulting with your Eye Gare Professional
- Always follow directions in the package inserts for the use of contact lens solutions. Use only a chemical (not heat) lens care system. Use of a heat (the mail care
- system can damage these lenses Staff aun preserved solutions, when used, should be discarded after the time specified in the disc stons.
- Do not use salita or anything other than the recommended solutions for lubit cating or welling lesses.
- Always is eap in sienses completely immersed in the ecommended storage solution when the lenses are not being worn glored; Prolonged periods of drying will reduce the solid light eleministration of results of drying will reduce the solid light eleministration of results. Follow the lens came directions in 'Case For A Dried Out (Dehydrated) Larti' films stuff and does become died out.

### r Topic a to Discuss with Patients:

- Always contact the Eve Care Professional before using any medicine in the
- eyes. Oratin medications, such as an thisterine a, decongestants, duellos, muscle relaxants, tanequillers, and those for motion sideness may cause dynams of the eye, horseased lens assertess, or bits of violent bands on millions exist, proper remedial measures should be peoples (Deprint growth passes). If the oxide high delivers of bands and people in this we highlight for use with not fortical lenses or the temprany discontinuation of ortical terms are writes and medication being used.
- Oral contraceptive users could develop visual changes or changes in lens tolerance when using contact, lenses. Palents should be caution accordingly.
- As with any contact, lens, follow-up visits are necessary to assure the con-tinuing heal h of the patient's eyes. The patient should be instructed as to a recommended follow-up schedule.

### Who Should Know That the Patient is Wearing Contact Lenses?

- Patients should inform all dioctors (Health Gare Professionals) about being
- Patients should always into mitheir employer of being a contact, lens wearer. Some jobs may require use of eye protection equipment or may require that the patient not wear contact lenses.

other eye disorders. The Bye Care Professional should be consulted for

### INDICATIONS (USES)

The ACUALE CASTS\* Brand Contact, Lenn is indicated for the optical correction of rethat/harmetropia (ryopia and hype opin) in phasic or aphalop a sons with non-diseased eyes who have 100 or less of additional formation. The ACUALE CASTS\* Brand Contact, Lenn for ASTGMATISM is indicated for the

These terres own.

Living and the third present of the system of the present of t requently isnned replacement was, the leasing a chemical disinfection system only.

targ at overhead underson agreem on the first specific of daily and extended wear for up to Brightar? days of continuous wear. It is recommended that, the contact lens wearer first the evaluated on a daily wear and wide. All suppose that, then a gradual introduction of extended wear can be followed as determined by the pie surfling Eye Claim.

These lenses are also indicated for therapeutic use as a banda geliens for the follow-

- For commany protection in Islands comeal almo mallises such as ent. opion, trichissis, tansal scara, and recurrent comeal existen. In addition, they are indicated for protection where solutions or opia structus emailorandism, degeneration or planships may result, in the need to protect the comes from explosure or repeated intaction.
- For use as a bar led du ing the healing process of epithelial de fects such as chronicegh in halls defects, comest does neuro topics and neuro paralytic learning, and chemical burns.

  For post surgicial confidirs survives bands ge lens use is indicated such as post refractive surgery, lametar g also, come all flags, and additional couler.

### ADVERSE REACTIONS

- There may be less comfort than when the lens was first placed on the eye.
- . There may be a feeling of something in the eye (foreign body, scratched There may be the potential for some temporary impairment due to
- I meetining die trieg poorties projekt eigengen zijn gegen die de projekt en de projek
- There may be expective wide that unusual eve permetions or surfaces of Poor visual aculty blurred vision, rain bows or halo s around objects, photo-
- phobia, or dry eyes may also o ocur if the lenses are worn continuously or
- The patient should be instructed to conduct a simple 8-part self-examina-tion at least once a day. They should ask themselves:
- How do the lenses feel on my eyes?
   How do my eyes look?
   Have In offced a change in my usen?
- If the patient reports any problems, he or she should be instructed to MIMEDIATE-

D/REMOVETHE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new fesh lens on the eye. If after in setting the new lens, the problem continues, the patient should be dreded to INMEDIATELY REMOVETHELENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL.

The patient should be instructed NOT to use an ewiens as self-treatment for the

setious condition such as infection, comeal ulos; necrossociarization or initis may be present. He or she should be instructed to seek immediate policional identifi-cation of the problem and prompt to atment to avoid serious eye diamage.

For structural stability and protection in pig gy back lens fitting where the cor-nea and associated surfaces are too irregular to allow for co-neal jigd gas permasa in (GPI) lenses to be it. In addition, thus so of the instruction prevent, initiation and abtrasions in conditions where the earse elevation differences in the hostig any junction or scar fasture.

prescribed for therapeutic use may be worn for dially or extended wearing

### CONTRAINDICATIONS (REASONS NOT TO USE)

- . As ale or subscute inflammation or infection of the anterior chamber of the
- Any eye disease, in jury or abnormality that affects the comes, conjunctiva
- Sa vere insufficien cy of iscrimal secretion (dry eye) Comes homosothesis ( adipadi comes) sensith M

- gerated by weating contact, sense or use or contact, the sections set of Coular install on due to allege reactions which may be caused by use of contact, lens solutions (a., cleaning and disinfecting solutions, rewelting drops, etc.) that contain chemicals or preserval was study as on a surport Thimerosal, all of to which so map explaining develop an allergic supprise.
- Any active comeal infection (black tail, fungal, protozoal or shall) · l'eyes become red or ir listed

For THERAPELITIC USE, the Eye Gare Professional may prescribe these lenses to add in the healing process of certain coular conditions, which may include those cited above.

Patients should be advised of the following warnings pertaining to contact lens wear:

EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAP DLY AND LEAD TO LOSS OF WISION; IF THE PATIENT EXPERIENCES:

### GENERAL FITTING GUIDELINES

### Patient Selection: Patients selected to wear these lenses should be chosen based on:

- Motivation to wear lenses Ability to follow instructions: a garding lens wear care
- Uservirsa recest
   Ability to adequately handle and care for the lenses
   Ability to understand the risk and benefits of lens wear
- Patients who do not meet the above criter's should not be provided with

Plaifiest who do not meet this above orest a amouse not per process must contract interest of the plain of the patient should be ginwth althorough case history to determine if there are any contain faction to contact here were. During the case history, the patient's value makes and expectation should be determined as well as an assessment of their overall could be physical, and mental health Preceding the initial selection of trial contact lenses, a comprehensive ocular evaluation should be performed that includes, but is not limited to, the mea-

surement of distance and near visual acuity, distance and near refractive pre-scription (notuding determining their elemed reading distance for presbyopes) Based on this evaluation, if it is determined that the platent is eligible to wear these lenses, it of the Care Professional should proped to the appropriate lens fitting lost up to a cultimate hallow.

C. In tail Power Betermination
A spectacle refs of on should be performed to establish the patent's baseline
ref active status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refis of on is gleater than a4.000.

Base & Curve Selection (final Lens Fitting)
The following trial lenses should be selected for patients regardless of leastorm by readings. However, corneal curvature measurements should be performed treatable the patient's baseline out tentature.

The trial lenses should be placed one ach of the patient's eyes and evaluated after the patient has adjusted to the lenses.

· ACUVUE GASYS\*: 84 mm/14.0 mm ACUVUE OASYS\* for ASTIGMATISM: 8.6mm/1.46 mm ACUVUE OASYS\* for PRESSYOP A: 8.4 mm/1.43 mm

- · Or Other BrePro

### THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY REM LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESSIO When prescribed for daily wear, patients should be instructed not to wear lenses while sleeping. Glinical studies have shown that the risk of sellows advance another is to be accorded to the lenses are some as the public and that it.

- Studies have shown that contact lens wearers who are smoke shave a higher incidence of adverse—eactions than nonsmokers.
- Problems with contact lenses or lens care products could result in setous injury to the eye. Patients should be cautioned that proper use and care of contact. enses and lens care products, in cluding lens cases, are essential for the safe are of these products.

Jare, in cluding cleaning the rest custom. didne, September 21, 1989, 931 (U), pp. 779-789

### Specific hatructions for Use and Warnings:

Instructions for Use

Wither can harbor microorganisms that can lead to sewere infection, vision loss or bindwiss. If items have been submessed in suder when participathy in water spectra or setterning in pools, in this can, bises or cossum, the palent should be intuitive to discard them and replace them with an every pair. The Tigs Case Professional should be consulted for commendations agarding watering intense to the commendation of the commendations.

during any activity in volving water · Soaking and Storing Your Lenger

ntact lens dish fecting) solution each time the

lenses are soaked (stored) The not reuse or "top off" of a solution left in the lens case since solution reuse educes effective lens disinfection and oo uid lead to se were infection, vision loss; or b lindh east.

1. Criteria of a Procedy F1 Lena A properly it lens will omite and completely cover the comes (i.e., no limbal accounts) in the contract file provide lear acchange under the contract lens with the birds, and to a control table. The term should move freely when manipulated display with in allower (iii, and then return to late power) contraved.

2. Citaria of a Fist Filtra Lane.
A fast filting lens may exhibit one or more of the following charactel stico: decentration, he complete command coverage (i.e., i intelli exposul e) exceeds wowment with the blink and/or edge standoff if the lens is judged to be fifs fitting, it should not be diagramed to the patient.

sleep fiting, it should not be dispensed to the patient.

8. Gilaria of a Steep Fitting Lera: Auteen fitting lerar may adhib to no or more of the 50 loveling characteristics: Insulficient movement with the blink; continue total indentation, and resistance when pushing the ien aup digitally with the lower list if the lerar is judged dis be

If the initial trial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the platient has adjusted to the lens: The lens should move feely when manipulated digitally with lower lid, and then return to an openity centered position when missioned. If resistance is encountered when pushing the lens up, the lens is fiting tightly and should not be dispensed to the patient.

Diagnosticiens

A spherical own e-shadon should be performed to determine the final i-power after the lens fit is judged acceptable. The appearable should be owner-estable should be combined with the trial lens power to determine the final lens scription. The patient should expe lense good visual acusty with the com-

+0.25D

| a description is anywers a second and a second contract of | |
|------------------------------------------------------------|--------|
| ample 1 | |
| agnostic lens: | -2 000 |
| herical over-refraction: | -0 250 |
| ral lens power: | -2 25D |

JJVC CONFIDENTIAL CR-6100, v 2.0 Page 81 of 117

# **APPENDIX D:**

| Lens Fitting Characteristics |
|---------------------------------------------------------|
| Subject Reported Ocular Symptoms/Problems |
| Determination of Distance Spherocylindrical Refractions |
| Biomicroscopy Scale |
| Distance and Near Visual Acuity Evaluation |
| Patient Reported Outcomes |

# LENS FITTING CHARACTERISTICS















# SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS



# DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS


















# **BIOMICROSCOPY SCALE**















# DISTANCE AND NEAR VISUAL ACUITY EVALUATION












# PATIENT REPORTED OUTCOMES



# APPENDIX E: DETERMINATION OF EYE DOMINANCY

# **+1.00 D LENS TEST**

| Step | Procedure |
|---|---|
| 1 | Place the subjects best sphero-cylindrical distance refraction in a trial frame |
| 2 | Have the subject view a BVA line of letters |
| 3 | With both eyes open alternate a +1.00 D trial lens between the right and left eye and ask the subject to indicate over which eye does the lens cause the line of letters to appear more blurred. The eye that the greatest blur is reported is the distance dominant eye. If the subject indicates that the amount of blur is about the same between the two eyes then record as neither eye dominant. |

# SIGHTING OCULAR DOMINANCE

| Step | Procedure |
|---|---|
| 1 | Ask the subject to extend both arms out and use his/her hands to form a triangle. The subject will be asked to keep both eyes open, and look through the triangle at a small object on the wall (e.g., a light switch or doorknob). |
| 2 | <ul> <li>Occlude the subject's left eye, then right eye. While alternating the occluder from the subject's eyes, ask the subject when they see the object.</li> <li>A. If the subject sees the object when the left eye is covered, the subject is <i>right eye</i> dominant.</li> <li>B. If the subject sees the object when the right eye is covered, the subject is <i>left eye</i> dominant.</li> <li>C. If the subject sees the object with both eyes, the opening between the hands may be too large. Therefore, ask the subject to make a smaller opening and repeat the procedure</li> </ul> |

# **APPENDIX F: IRIS COLOR**



# APPENDIX G: SPECTRUM OF THE UV ACTUATOR



# APPENDIX H: STARBURST AND HALO IMAGES







# PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6100 The effects of contact lenses with experimental dye on visual function

Version and Date: v2.0 07 June 2018

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |